CLINICAL TRIAL: NCT02008227
Title: A Phase III, Open-Label, Multicenter, Randomized Study to Investigate the Efficacy and Safety of Atezolizumab (Anti-PD-L1 Antibody) Compared With Docetaxel in Patients With Non-Small Cell Lung Cancer After Failure With Platinum Containing Chemotherapy
Brief Title: A Study of Atezolizumab Compared With Docetaxel in Participants With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Who Have Failed Platinum-Containing Therapy
Acronym: OAK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO28915; 2013-003331-30 (EudraCT Number)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — atezolizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody (Experimental): Atezolizumab 1200 milligrams (mg) was administered via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression, death, unacceptable toxicity, withdrawal of consent, or study termination by sponsor, whichever occurs first.
  Interventions: Drug: Atezolizumab
- Docetaxel (Active Comparator): Docetaxel 75 milligrams per meter square (mg/m^2) was administered via IV infusion on Day 1 of each 21-day cycle until disease progression, death, unacceptable toxicity, withdrawal of consent, or study termination by sponsor, whichever occurs first.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg IV infusion on Day 1 of each 21-day cycle
  Other Names: Tecentriq
  Arms: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
Drug: Docetaxel — 75 mg/m^2 IV infusion on Day 1 of each 21-day cycle
  Arms: Docetaxel

SUMMARY:
This global, multicenter, open-label, randomized, controlled study evaluated the efficacy and safety of atezolizumab (an anti-programmed death-ligand 1 [anti-PD-L1] antibody)compared with docetaxel in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) after failure with platinum-containing chemotherapy. Participants were randomized 1:1 to receive either docetaxel or atezolizumab. Treatment may continue as long as participants experienced clinical benefit as assessed by the investigator, i.e., in the absence of unacceptable toxicity or symptomatic deterioration attributed to disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic (Stage IIIB, Stage IV, or recurrent) NSCLC
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens
* Disease progression during or following treatment with a prior platinum-containing regimen for locally advanced, unresectable/inoperable or metastatic NSCLC or disease recurrence within 6 months of treatment with a platinum-based adjuvant/neoadjuvant regimen or combined modality (e.g., chemoradiation) regimen with curative intent
* Measurable disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Known active or untreated central nervous system (CNS) metastases
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Active hepatitis B or hepatitis C
* Prior treatment with docetaxel
* Prior treatment with cluster of differentiation 137 (CD137) agonists, anti-cytotoxic-T-lymphocyte-associated antigen 4 (anti-CTLA4), anti-programmed death-1 (anti-PD-1), or anti-PD-L1 therapeutic antibody or pathway-targeting agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1225 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2016-07-07 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (208):
- United States (59):
  - Comprehensive Blood/Cancer Ctr, Bakersfield, California
  - Roy & Patricia Disney Family Cancer Center, Burbank, California
  - St. Jude Heritage Healthcare; Virgiia K.Crosson Can Ctr, Fullerton, California
  - Kaiser Permanente - Hayward, Hayward, California
  - Scripps Clinic; Hematology & Oncology, La Jolla, California
  - Pacific Shores Medical Group, Long Beach, California
  - Univ of Calif, Los Angeles; Hematology/Oncology, Los Angeles, California
  - North Valley Hem Onc Med Grp; Thomas&Dorothy Leavey Can Ctr, Northridge, California
  - Kaiser Permanente - Oakland, Oakland, California
  - TMPN/ Cancer Care Associates, Redondo Beach, California
  - Kaiser Permanente - Roseville, Roseville, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - UC Davis; Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente - San Francisco (2238 Geary), San Francisco, California
  - K. Permanente - San Jose, San Jose, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Kaiser Permanente - San Marcos, San Marcos, California
  - K. Permanente - Santa Clara, Santa Clara, California
  - Central Coast Medical Oncology, Santa Maria, California
  - K. Permanente - S. San Fran, South San Francisco, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - K. Permanente - Walnut Creek, Walnut Creek, California
  - St. Mary's Hospital Regional Cancer Center, Grand Junction, Colorado
  - Kaiser Permanente - Franklin; Kaiser Permanente - Lone Tree, Lone Tree, Colorado
  - Cancer Specialists; North Florida ;Jacksonville (AC Skinner Pkwy), Jacksonville, Florida
  - AMPM Research Clinic, Miami, Florida
  - Orlando Health Inc., Orlando, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Hematology-Oncology; Associates of the Quad Cities, Bettendorf, Iowa
  - New England Cancer Specialists, Scarborough, Maine
  - Karmanos Cancer Inst. ; Hudson Webber; Cancer Research Building, Detroit, Michigan
  - US Oncology Research at Minnesota Oncology, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Billings Clinic; Research Center, Billings, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Oncology Hematology West Midwest, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Eastern Avenue, Las Vegas, Nevada
  - Summit Medical Center, Florham Park, New Jersey
  - Luckow Pavillion, Valley Hosp; Office of Clinical Trials, Paramus, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Roswell Park Cancer Inst., Buffalo, New York
  - New York Oncology Hematology PC - Latham, Clifton Park, New York
  - Mid Ohio Onc Hematology Inc, Columbus, Ohio
  - Cancer Treatment Centers of America-Tulsa, Tulsa, Oklahoma
  - Willamette Valley Cancer Ctr - 520 Country Club, Eugene, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Texas Onc-Central Austin CA Ct, Austin, Texas
  - The Methodist Cancer Center, Houston, Texas
  - Texas Oncology, P.A. - Tyler; Tyler Cancer Center, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
  - Aurora Health Care; Patient Centered Research, Milwaukee, Wisconsin
- Argentina (3):
  - Instituto Medico Rio Cuarto, Córdoba
  - COIBA, Provincia de Buenos Aires
  - Instituto de Oncología de Rosario, Rosario
- Austria (3):
  - Lkh innsbruck - univ. Klinikum innsbruck - Tiroler landeskrankenanstalten ges.m.b.h.; Innere Medizin, Innsbruck
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - Lkh Vöcklabruck; I. Abt. Für Innere Medizin, Vöcklabruck
- Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Cite de La Sante de Laval; Hemato-Oncologie, Laval, Quebec
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
- Chile (3):
  - Bradford Hill Centro de Investigaciones Clinicas; Bradford Hill Centro de Investigaciones Clinicas, Recoleta
  - Sociedad de Investigaciones Medicas Ltda (SIM), Temuco
  - ONCOCENTRO APYS; Oncología, Viña del Mar
- Finland (3):
  - Helsinki University Central Hospital; Dep. of Pulmonary Medicine, Helsinki
  - Oulu University Hospital; Oncology, Oulu
  - Tampere University Hospital; Dept of Oncology, Tampere
- France (21):
  - Institut Sainte Catherine, Avignon
  - Hopital Jean Minjoz; Pneumologie, Besançon
  - Polyclinique Bordeaux Nord Aquitaine; Chimiotherapie Radiotherapie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier Intercommunal; Service de Pneumologie, Créteil
  - Chu Grenoble - Hopital Albert Michallon; Departement de Cancero-Hematologie, Grenoble
  - Centre Jean Bernard; Radiotherapie Chimiotherapie, Le Mans
  - Centre Oscar Lambret, Lille
  - Hopital Nord; Service d'Oncologie Multidisciplinaire et Innovation Thérapeutique, Marseille
  - Hopital Emile Muller;Pneumologie, Mulhouse
  - Hopital Cochin; Unite Fonctionnelle D Oncologie, Paris
  - Hopital Saint Louis; Oncologie Medicale, Paris
  - GH Paris Saint Joseph; Pneumologie, Paris
  - Hopital Tenon;Pneumologie, Paris
  - Centre Hospitalier Lyon Sud; Pneumologie, Pierre-Bénite
  - CH de la region d Annecy, Pringy
  - Hopital de Pontchaillou; Service de Pneumologie, Rennes
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Hopital Foch; Pneumologie, Suresnes
  - Hia Sainte Anne; Pneumologie, Toulon
  - Hopital Larrey; Pneumologie, Toulouse
- Germany (9):
  - Helios Klinikum Emil von Behring GmbH, Berlin
  - Krankenhaus Merheim Lungenklinik, Cologne
  - Krankenhaus Nordwest; Klinik f. Onkologie und Hämatologie, Frankfurt
  - Asklepios-Fachkliniken Muenchen-Gauting; Onkologie, Gauting
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH; Klinik fuer Innere Medizin II, Halle
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - Universitätsklinikum Regensburg; Klinik und Poliklinik für Innere Medizin II, Pneumologie, Regensburg
- Greece (3):
  - Uoa Sotiria Hospital; Oncology, Athens
  - University Hospital of Patras Medical Oncology, Pátrai
  - Thermi Clinic; Oncology Clinic, Thermi Thessalonikis
- Grupo Angeles, Guatemala City, Guatemala
- Hungary (3):
  - Semmelweis Egyetem X; Pulmonologiai Klinika, Budapest
  - University of Pecs, I st Dept of Internal Medicine, Pécs
  - Tudogyogyintezet Torokbalint, Törökbálint
- Italy (16):
  - Irccs Ist. Tumori Giovanni Paolo Ii; Dipartimento Oncologia Medica, Bari, Apulia
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino, Campania
  - Seconda Universita' Degli Studi; Divsione Di Oncologia Medica, Napoli, Campania
  - Azienda Ospedaliera Univ Parma; Dept Oncologia Medica, Parma, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - Azienda Ospedaliero-Uni Ria Di Udine; Dept. Di Oncologia - Padiglione Pennato, Udine, Friuli Venezia Giulia
  - Uni Cattolica Policlinico Gemelli; Oncologia Medica Ist. Medicina Interna, Rome, Lazio
  - Istituto Nazionale per la Ricerca sul Cancro di Genova, Genoa, Liguria
  - Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - ASST DI MONZA; Oncologia Medica, Monza, Lombardy
  - POLICLINICO RODOLICO, U.O. di Oncologia Medica, Catania, Sicily
  - Ospedale San Luca; Oncologia, Lucca, Tuscany
  - A.O. Universitaria Pisana-Ospedale Cisanello; Dipartimento Cardio Toracico-Pneumologia Ii, Pisa, Tuscany
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Seconda, Padua, Veneto
  - A.O.U. Integrata Verona - Policlinico G.B. Rossi; Oncologia Medica - Dip. di Medicina, Verona, Veneto
- Japan (16):
  - Aichi Cancer Center Hospital; Respiratory Medicine, Aichi
  - National Cancer Center Hospital East; Thoracic Oncology, Chiba
  - National Hospital Organization Shikoku Cancer Center; Internal Medicine, Ehime
  - National Hospital Organization Kyushu Cancer Center, Thoracic Oncology, Fukuoka
  - Kobe City Medical Center General Hospital; Respiratory Medicine, Hyōgo
  - Hyogo Cancer Center; Thoracic Oncology, Hyōgo
  - Miyagi Cancer Center; Respiratory Medicine, Miyagi
  - Okayama University Hospital; Respiratory and Allergy Medicine, Okayama
  - Kindai University Hospital; Medical Oncology, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center; Internal Medicine, Osaka
  - Saitama Cancer Center; Thoracic Oncology, Saitama
  - Shizuoka Cancer Center; Thoracic Oncology, Shizuoka
  - National Cancer Center Hospital; Thoracic Medical Oncology, Tokyo
  - The Cancer Institute Hospital of JFCR, Respiratory Medicine, Tokyo
  - Tokyo Medical University Hospital; Dept of Surgery, Tokyo
  - National Hospital Organization, Yamaguchi - Ube Medical Center; Oncology Medicine, Yamaguchi
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Catharina Ziekenhuis; Dept of Lung Diseases, Eindhoven
  - Antonius Ziekenhuis; Dept of Lung Diseases, Nieuwegein
- New Zealand (3):
  - Auckland city hospital; Auckland Regional Cancer Centre and Blood Service, Auckland
  - Dunedin Hospital, Dunedin
  - Waikato Hospital; Dept of Medical Oncology, Hamilton
- Oslo Universitetssykehus HF; Radiumhospitalet, Oslo, Norway
- Centro Hemato Oncologico Panama, Panama City, Panama
- Poland (5):
  - Medical University of Gdansk, Gdansk
  - Woj.Wielospecjalistyczne Centrum Onkologii i Traumatologii; Oddz.Hematologii Pododz.Chemioterapii, Lodz
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy; Oddzial Iii, Otwock
  - Med.-Polonia Sp. z o.o. NSZOZ, Poznan
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie Klinika Nowotworów Piersi i Chirurgii, Warsaw
- Portugal (3):
  - Hospital Geral; Servico de Pneumologia, Coimbra
  - Hospital Pulido Valente; Servico de Pneumologia, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Russia (3):
  - N.N.Burdenko Main Military Clinical Hospital; Oncology Dept, Moscow
  - City Clinical Onc., Saint Petersburg
  - SBI of Healthcare Samara Regional Clinical Oncology Dispensary, Samara
- Serbia (2):
  - Clinic for Pulmonology, Clinical Center of Serbia, Belgrade
  - Institute for pulmonary diseases of Vojvodina, Kamenitz
- South Korea (6):
  - National Cancer Center; Medical Oncology, Gyeonggi-do
  - Seoul National University Bundang Hospital; Hematology Medical Oncology, Gyeonggi-do
  - Seoul National Uni Hospital; Internal Medicine, Seoul
  - Yonsei University Severance Hospital; Medical Oncology, Seoul
  - Samsung Medical Center; Gastroenterology, Seoul
  - Seoul St.Mary's Hospital; Medical Oncology, Seoul
- Spain (10):
  - Hospital Universitario Materno Infantil de Gran Canaria; Servicio de Oncologia, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario Puerta de Hierro; Servicio de Oncologia, Majadahonda, Madrid
  - Complejo Hospitalario Universitario A Coruña (CHUAC, Materno Infantil), Oncología, A Coruña
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Fundacion Jimenez Diaz; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Oncologia, Málaga
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Lungmedicinkliniken, Gothenburg
  - Universitetssjukhuset Linköping; Lungmedicinkliniken, Linköping
  - Karolinska Universitetssjukhuset, Solna; Lung Allergikliniken N10:02, Stockholm
- Switzerland (3):
  - Kantonsspital Baden; Medizinische Klinik, Onkologie, Baden
  - HUG; Oncologie, Geneva
  - Luzerner Kantonsspital; Medizinische Onkologie, Lucerne
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Taiwan Uni Hospital; Internal Medicine, Taipei
  - Taipei Veterans General Hospital; Chest Dept , Section of Thoracic Oncology, Taipei
  - Chang Gung Medical Foundation - Linkou; Division of Hematology- Oncology, Taoyuan District
- Thailand (3):
  - Chulalongkorn Hospital; Medical Oncology, Bangkok
  - Ramathibodi Hospital; Dept of Med.-Div. of Med. Onc, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
- Turkey (Türkiye) (2):
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital; Medical Oncology, Istanbul
  - Izmir Suat Seren Chest Diseases and Surgery Research Hospital, Izmir
- Ukraine (3):
  - State Medical Academy; Oncology, Dnipropetrovsk
  - Karkiv Regional Oncology Center, Kharkiv
  - Uzhgorod Nat. University Central Municip Hosp; Onc Center, Uzhhorod
- United Kingdom (8):
  - Diana Princess of Wales Hosp., Grimsby
  - University College London Hospital, London
  - Royal Free Hospital, London
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - St George's Hospital, London
  - Charing Cross Hospital, London
  - Christie Hospital NHS Trust, Manchester
  - Kings Mill Hospital, Sutton in Ashfield

REFERENCES:
- [Derived] Melchionna R, Di Modugno F, Di Carlo A, D'Ambrosio L, Palermo B, Tocci A, Paolini F, Sperduti I, Campo G, Taje R, Gallina F, Visca P, D'Andrea D, Nistico P. Reciprocal regulation of hMENA and TGF-beta signaling in cancer-associated fibroblasts promotes EMT, immunosuppression, poor prognosis, and ICT resistance in NSCLC. J Immunother Cancer. 2026 Jan 27;14(1):e013098. doi: 10.1136/jitc-2025-013098. PMID 41592891
- [Derived] Mhatre SK, Machado RJM, Ton TGN, Trinh H, Mazieres J, Rittmeyer A, Bretscher MT. Real-World Progression-Free Survival as an Endpoint in Lung Cancer: Replicating Atezolizumab and Docetaxel Arms of the OAK Trial Using Real-World Data. Clin Pharmacol Ther. 2023 Dec;114(6):1313-1322. doi: 10.1002/cpt.3045. Epub 2023 Sep 28. PMID 37696652
- [Derived] Saal J, Bald T, Eckstein M, Ritter M, Brossart P, Ellinger J, Holzel M, Klumper N. Early C-reactive protein kinetics predicts immunotherapy response in non-small cell lung cancer in the phase III OAK trial. JNCI Cancer Spectr. 2023 Mar 1;7(2):pkad027. doi: 10.1093/jncics/pkad027. PMID 37004206
- [Derived] Dong Y, Zhu Y, Zhuo M, Chen X, Xie Y, Duan J, Bai H, Hao S, Yu Z, Yi Y, Guan Y, Yuan J, Xia X, Yi X, Wang J, Wang Z. Maximum Somatic Allele Frequency-Adjusted Blood-Based Tumor Mutational Burden Predicts the Efficacy of Immune Checkpoint Inhibitors in Advanced Non-Small Cell Lung Cancer. Cancers (Basel). 2022 Nov 17;14(22):5649. doi: 10.3390/cancers14225649. PMID 36428744
- [Derived] Cortellini A, Ricciuti B, Borghaei H, Naqash AR, D'Alessio A, Fulgenzi CAM, Addeo A, Banna GL, Pinato DJ. Differential prognostic effect of systemic inflammation in patients with non-small cell lung cancer treated with immunotherapy or chemotherapy: A post hoc analysis of the phase 3 OAK trial. Cancer. 2022 Aug 15;128(16):3067-3079. doi: 10.1002/cncr.34348. Epub 2022 Jun 21. PMID 35727053
- [Derived] Gadgeel S, Hirsch FR, Kerr K, Barlesi F, Park K, Rittmeyer A, Zou W, Bhatia N, Koeppen H, Paul SM, Shames D, Yi J, Matheny C, Ballinger M, McCleland M, Gandara DR. Comparison of SP142 and 22C3 Immunohistochemistry PD-L1 Assays for Clinical Efficacy of Atezolizumab in Non-Small Cell Lung Cancer: Results From the Randomized OAK Trial. Clin Lung Cancer. 2022 Jan;23(1):21-33. doi: 10.1016/j.cllc.2021.05.007. Epub 2021 May 30. PMID 34226144
- [Derived] Gandara D, Reck M, Moro-Sibilot D, Mazieres J, Gadgeel S, Morris S, Cardona A, Mendus D, Ballinger M, Rittmeyer A, Peters S. Fast progression in non-small cell lung cancer: results from the randomized phase III OAK study evaluating second-line atezolizumab versus docetaxel. J Immunother Cancer. 2021 Mar;9(3):e001882. doi: 10.1136/jitc-2020-001882. PMID 33737340
- [Derived] Shemesh CS, Chan P, Legrand FA, Shames DS, Das Thakur M, Shi J, Bailey L, Vadhavkar S, He X, Zhang W, Bruno R. Pan-cancer population pharmacokinetics and exposure-safety and -efficacy analyses of atezolizumab in patients with high tumor mutational burden. Pharmacol Res Perspect. 2020 Dec;8(6):e00685. doi: 10.1002/prp2.685. PMID 33241650
- [Derived] Chalabi M, Cardona A, Nagarkar DR, Dhawahir Scala A, Gandara DR, Rittmeyer A, Albert ML, Powles T, Kok M, Herrera FG; imCORE working group of early career investigators. Efficacy of chemotherapy and atezolizumab in patients with non-small-cell lung cancer receiving antibiotics and proton pump inhibitors: pooled post hoc analyses of the OAK and POPLAR trials. Ann Oncol. 2020 Apr;31(4):525-531. doi: 10.1016/j.annonc.2020.01.006. Epub 2020 Jan 16. PMID 32115349
- [Derived] Morrissey KM, Marchand M, Patel H, Zhang R, Wu B, Phyllis Chan H, Mecke A, Girish S, Jin JY, Winter HR, Bruno R. Alternative dosing regimens for atezolizumab: an example of model-informed drug development in the postmarketing setting. Cancer Chemother Pharmacol. 2019 Dec;84(6):1257-1267. doi: 10.1007/s00280-019-03954-8. Epub 2019 Sep 21. PMID 31542806
- [Derived] Gadgeel SM, Lukas RV, Goldschmidt J, Conkling P, Park K, Cortinovis D, de Marinis F, Rittmeyer A, Patel JD, von Pawel J, O'Hear C, Lai C, Hu S, Ballinger M, Sandler A, Gandhi M, Fehrenbacher L. Atezolizumab in patients with advanced non-small cell lung cancer and history of asymptomatic, treated brain metastases: Exploratory analyses of the phase III OAK study. Lung Cancer. 2019 Feb;128:105-112. doi: 10.1016/j.lungcan.2018.12.017. Epub 2018 Dec 19. PMID 30642441
- [Derived] Bordoni R, Ciardiello F, von Pawel J, Cortinovis D, Karagiannis T, Ballinger M, Sandler A, Yu W, He P, Matheny C, Felizzi F, Rittmeyer A. Patient-Reported Outcomes in OAK: A Phase III Study of Atezolizumab Versus Docetaxel in Advanced Non-Small-cell Lung Cancer. Clin Lung Cancer. 2018 Sep;19(5):441-449.e4. doi: 10.1016/j.cllc.2018.05.011. Epub 2018 May 31. PMID 30017645
- [Derived] Hida T, Kaji R, Satouchi M, Ikeda N, Horiike A, Nokihara H, Seto T, Kawakami T, Nakagawa S, Kubo T. Atezolizumab in Japanese Patients With Previously Treated Advanced Non-Small-Cell Lung Cancer: A Subgroup Analysis of the Phase 3 OAK Study. Clin Lung Cancer. 2018 Jul;19(4):e405-e415. doi: 10.1016/j.cllc.2018.01.004. Epub 2018 Feb 1. PMID 29525239
- [Derived] Rittmeyer A, Barlesi F, Waterkamp D, Park K, Ciardiello F, von Pawel J, Gadgeel SM, Hida T, Kowalski DM, Dols MC, Cortinovis DL, Leach J, Polikoff J, Barrios C, Kabbinavar F, Frontera OA, De Marinis F, Turna H, Lee JS, Ballinger M, Kowanetz M, He P, Chen DS, Sandler A, Gandara DR; OAK Study Group. Atezolizumab versus docetaxel in patients with previously treated non-small-cell lung cancer (OAK): a phase 3, open-label, multicentre randomised controlled trial. Lancet. 2017 Jan 21;389(10066):255-265. doi: 10.1016/S0140-6736(16)32517-X. Epub 2016 Dec 13. PMID 27979383

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twelve hundred and twenty-five participants were randomized in the study and were considered the Secondary Population (SP), out of which first 850 randomized participants were considered the Primary Population (PP).
Groups:
- Docetaxel: Docetaxel 75 milligrams per square meter (mg/m^2) was administered intravenously (IV) on Day 1 of each 21-day cycle until disease progression, death, unacceptable toxicity, withdrawal of consent, or study termination by sponsor, whichever occurred first.
- Atezolizumab: Atezolizumab 1200 milligrams (mg) was administered IV on Day 1 of each 21-day cycle until disease progression or loss of clinical benefit, death, unacceptable toxicity, withdrawal of consent, or study termination by sponsor, whichever occurred first.
Period: Overall Study
Arm/Group | Docetaxel | Atezolizumab
Started | 612 | 613
Treated | 579 | 608
Completed | 0 | 0
Not Completed | 612 | 613
Not completed — Lost to Follow-up | 7 | 9
Not completed — Death | 494 | 485
Not completed — Withdrawal by Subject | 67 | 36
Not completed — Study Terminated By Sponsor | 44 | 83

BASELINE CHARACTERISTICS:
Population: SP-Intent to Treat (ITT) analysis set included all randomized ITT participants regardless of whether they received any study drug.
Groups:
- Atezolizumab: Atezolizumab 1200 mg was administered IV on Day 1 of each 21-day cycle until disease progression or loss of clinical benefit, death, unacceptable toxicity, withdrawal of consent, or study termination by sponsor, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Docetaxel | Atezolizumab | Total
Number analyzed (Participants) | 612 | 613 | 1225
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (9.2) | 62.7 (9.8) | 62.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 234 | 467
  Male | 379 | 379 | 758
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 48 | 90
  Not Hispanic or Latino | 541 | 540 | 1081
  Unknown or Not Reported | 29 | 25 | 54
Race/Ethnicity, Customized [Number; unit: Participants] — Population: SP-ITT Population
  Participants
    American Indian or Alaska Native: number analyzed (Participants) | 2 | 1 | 3
    American Indian or Alaska Native | 2 | 1 | 3
    Asian: number analyzed (Participants) | 125 | 124 | 249
    Asian | 125 | 124 | 249
    Black or African American: number analyzed (Participants) | 16 | 11 | 27
    Black or African American | 16 | 11 | 27
    Native Hawaiian or other Pacific Islander: number analyzed (Participants) | 2 | 3 | 5
    Native Hawaiian or other Pacific Islander | 2 | 3 | 5
    White: number analyzed (Participants) | 432 | 438 | 870
    White | 432 | 438 | 870
    Other: number analyzed (Participants) | 12 | 11 | 23
    Other | 12 | 11 | 23
    Multiple: number analyzed (Participants) | 1 | 2 | 3
    Multiple | 1 | 2 | 3
    Unknown: number analyzed (Participants) | 22 | 23 | 45
    Unknown | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Died: PP-ITT
Time Frame: Baseline until death due to any cause (up to approximately 2.25 years)
Population: PP-ITT analysis set included the first 850 randomized ITT participants regardless of whether they received any study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Percentage of Participants | 70.1 | 63.8

2. Primary Outcome: Percentage of Participants Who Died: Tumor Cells (TC)1/2/3 or Tumor-Infiltrating Immune Cells (IC)1/2/3 Subgroup of PP
Description: Percentage of participants who died among TC1/2/3 or IC1/2/3 subgroup of PP-ITT were reported. TC1 = presence of discernible programmed death-ligand 1 (PD-L1) staining of any intensity in >/=1% and <5% TCs; TC2: presence of discernible PD-L1 staining of any intensity in >/=5% and <50% TCs; TC3 = presence of discernible PD-L1 staining of any intensity in >/=50% TCs; IC1 = presence of discernible PD-L1 staining of any intensity in ICs covering between >/=1% and <5% of tumor area occupied by tumor cells, associated intratumoral, and contiguous peri-tumoral desmoplastic stroma; IC2 = presence of discernible PD-L1 staining of any intensity in ICs covering between >/=5% and <10% of tumor area occupied by tumor cells, associated intratumoral, and contiguous peri-tumoral desmoplastic stroma; IC3 = presence of discernible PD-L1 staining of any intensity in ICs covering >/=10% of tumor area occupied by tumor cells, associated intratumoral, and contiguous peri-tumoral desmoplastic stroma.
Time Frame: Baseline until death due to any cause (up to approximately 2.25 years)
Population: TC1/2/3 or IC1/2/3 subgroup within PP included ITT participants with the corresponding programmed death-ligand 1 (PD-L1) expression status.
Measure: Number; unit: Percentage of Participants
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 222 | 241
Percentage of Participants | 67.1 | 62.7

3. Primary Outcome: Overall Survival (OS): PP-ITT
Description: OS duration is defined as the difference in time from the date of randomization to the date of death due to any cause. Data for participants who were not reported as having died at the time of analysis were censored at the date they were last known to be alive. Participants who had no post-baseline information were censored at the date of randomization plus 1 day. OS was estimated using KM methodology.
Time Frame: Baseline until death due to any cause (up to approximately 2.25 years)
Population: The PP-ITT analysis set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Months | 9.6 [8.6 to 11.2] | 13.8 [11.8 to 15.7]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; Stratified analysis based on the strata of IC levels per interactive voice/web response system (IxRS), the number of prior chemotherapy regimens per IxRS, and histology per electronic case report form (eCRF); Test type: Superiority or Other; p = 0.0003, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.62 to 0.87]
Statistical Analysis 2: Comparison: Docetaxel vs Atezolizumab; Unstratified Analysis; Test type: Superiority or Other; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.62 to 0.86]

4. Primary Outcome: OS: TC1/2/3 or IC1/2/3 Subgroup of PP
Description: as for outcome 3
Time Frame: Baseline until death due to any cause (up to approximately 2.25 years)
Population: TC1/2/3 or IC1/2/3 subgroup of PP
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 222 | 241
Months | 10.3 [8.8 to 12.0] | 15.7 [12.6 to 18.0]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; Stratified analysis based on the strata of IC levels per IxRS, the number of prior chemotherapy regimens per IxRS, and histology per eCRF; Test type: Superiority or Other; p = 0.0102, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.58 to 0.93]
Statistical Analysis 2: Comparison: Docetaxel vs Atezolizumab; Unstratified Analysis; Test type: Superiority or Other; p = 0.0052, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.58 to 0.91]

5. Secondary Outcome: Percentage of Participants With Disease Progression (PD) as Determined by Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) or Death: PP-ITT
Description: PD: at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 millimeters (mm), or presence of new lesions.
Time Frame: Baseline up to PD or Death (up to approximately 2.25 years)
Population: The PP-ITT analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Percentage of Participants | 88.2 | 89.4

6. Secondary Outcome: Percentage of Participants With PD as Determined by Investigator Using RECIST v1.1 or Death: TC1/2/3 or IC1/2/3 Subgroup of PP
Description: PD: at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, or presence of new lesions.
Time Frame: Baseline up to PD or Death (up to approximately 2.25 years)
Population: TC1/2/3 or IC1/2/3 subgroup of PP
Measure: Number; unit: Percentage of Participants
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 222 | 241
Percentage of Participants | 86.9 | 89.6

7. Secondary Outcome: Progression-Free Survival (PFS) as Determined by Investigator Using RECIST v1.1: PP-ITT
Description: PFS is defined as the time between the date of randomization and the date of first documented PD or death, whichever occurs first. Participants who are alive and have not experienced PD at the time of analysis were censored at the time of the last tumor assessment. Participants with no post-baseline tumor assessment were censored at the randomization date plus 1 day. PD: at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, or presence of new lesions.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 2.25 years)
Population: The PP-ITT analysis set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Months | 4.0 [3.3 to 4.2] | 2.8 [2.6 to 3.0]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.4928, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.82 to 1.10]
Statistical Analysis 2: Comparison: Docetaxel vs Atezolizumab; Unstratified Analysis; Test type: Superiority or Other; p = 0.3596, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.81 to 1.08]

8. Secondary Outcome: PFS as Determined by Investigator Using RECIST v1.1: TC1/2/3 or IC1/2/3 Subgroup of PP
Description: as for outcome 7
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 2.25 years)
Population: The TC1/2/3 or IC1/2/3 subgroup of PP
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 222 | 241
Months | 4.1 [2.9 to 4.3] | 2.8 [2.6 to 4.0]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.3806, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.74 to 1.12]
Statistical Analysis 2: Comparison: Docetaxel vs Atezolizumab; Unstratified Analysis; Test type: Superiority or Other; p = 0.3249, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.74 to 1.10]

9. Secondary Outcome: Percentage of Participants With Objective Response as Determined Using RECIST v1.1: PP-ITT
Description: Objective response is defined as a complete response (CR) or partial response (PR) as determined by the Investigator using RECIST v1.1 on 2 consecutive occasions at least 6 weeks apart. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than [<] 10 mm). No new lesions. At least a 30% decrease in the sum of the diameters of all target and all new measurable lesions, taking as reference the baseline sum of diameters, in the absence of CR. No new lesions.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 2.25 years)
Population: The PP-ITT analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Percentage of Participants | 13.4 [10.32 to 17.02] | 13.6 [10.53 to 17.28]

10. Secondary Outcome: Percentage of Participants With Objective Response as Determined Using RECIST v1.1: TC1/2/3 or IC1/2/3 Subgroup of PP
Description: Objective response is defined as a CR or PR as determined by the Investigator using RECIST v1.1 on 2 consecutive occasions at least 6 weeks apart. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. At least a 30% decrease in the sum of the diameters of all target and all new measurable lesions, taking as reference the baseline sum of diameters, in the absence of CR. No new lesions.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 2.25 years)
Population: The TC1/2/3 or IC1/2/3 subgroup of PP
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 222 | 241
Percentage of Participants | 16.2 [11.62 to 21.74] | 17.8 [13.22 to 23.27]

11. Secondary Outcome: Duration of Response (DOR) as Determined by Investigator Using RECIST v1.1: PP-ITT
Description: DOR:Duration from the first tumor assessment that supports the participant's objective response to PD or death due to any cause,whichever occurs first.CR:complete disappearance of all target lesions and non-target disease.All nodes,both target and non-target,must decrease to normal. No new lesions.PR: At least a 30% decrease in the sum of the diameters of all target and all new measurable lesions, taking as reference the baseline sum of diameters, in the absence of CR.Participants who have not experienced PD at the time of analysis were censored at the time of the last tumor assessment.Participants with no post-baseline tumor assessment were censored at the randomization date plus 1 day.PD:at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm,progression of existing non-target lesions,or presence of new lesions.DOR was estimated using KM methodology.
Time Frame: From first objective response of CR or PR to PD or death due to any cause, whichever occurred first (up to approximately 2.25 years)
Population: The PP-ITT analysis set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 57 | 58
Months | 6.2 [4.9 to 7.6] | 16.3 [10.0 to NA] — Data not reported because the upper limit of confidence interval (CI) was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.18 to 0.55]
Statistical Analysis 2: Comparison: Docetaxel vs Atezolizumab; Unstratified Analysis; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.21 to 0.55]

12. Secondary Outcome: DOR as Determined by Investigator Using RECIST v1.1: TC1/2/3 or IC1/2/3 Subgroup of PP
Description: as for outcome 11
Time Frame: as for outcome 11
Population: The TC1/2/3 or IC1/2/3 subgroup of PP
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 36 | 43
Months | 6.2 [4.9 to 9.2] | 16.0 [9.7 to NA] — Data not reported because the upper limit of CI was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0006, Log Rank; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.15 to 0.62]
Statistical Analysis 2: Comparison: Docetaxel vs Atezolizumab; Unstratified Analysis; Test type: Superiority or Other; p = 0.0003, Log Rank; Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.22 to 0.65]

13. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) Against Atezolizumab
Time Frame: Baseline up to approximately 2.25 years (assessed at predose [Hour {Hr} 0] on Day 1 of Cycles 1, 2, 3, 4, 8, 16, then every 8 cycles up to end of treatment (EOT) [approximately 2.25 years]; 120 days after EOT [approximately 2.25 years] [1 Cycle=21 days])
Population: ATA evaluable population included all participants who received atezolizumab treatment and had at least one post treatment ATA result.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 565
Percentage of Participants | 30.4

14. Secondary Outcome: Maximum Observed Serum Atezolizumab Concentration (Cmax)
Time Frame: Predose (Hr 0), 30 minutes (min) post-infusion (infusion duration: 60 min) on Cycle 1 Day 1 (1 Cycle=21 days)
Population: Pharmacokinetic (PK) evaluable population included participants who received atezolizumab treatment and had at least one measurable PK concentration.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | Atezolizumab
Number analyzed (Participants) | 606
Microgram per milliliter (mcg/mL) | 400 (127)

15. Secondary Outcome: Minimum Observed Serum Atezolizumab Concentration (Cmin)
Time Frame: Predose (Hr 0) on Day 1 of Cycles 1, 2, 3, 4, 8, 16, 24, 32, EOT (approximately 2.25 years); 120 days after EOT (approximately 2.25 years) (1 Cycle=21 days)
Population: PK evaluable participants. Here, 'n' signifies those participants evaluated for this measure at specific time point. All 606 participants contributed to the endpoint but not all completed evaluation of every timepoint. Convention 'CxDx' refers to cycle number and day number.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab
Number analyzed (Participants) | 606
mcg/mL
  C1D1 (n= 593) | 2.59 (30.9)
  C2D1 (n= 534) | 83.2 (31.0)
  C3D1 (n= 445) | 130 (55.8)
  C4D1 (n= 405) | 158 (66.4)
  C8D1 (n= 222) | 205 (99.4)
  C16D1 (n= 132) | 226 (105)
  C24D1 (n= 63) | 250 (99.8)
  C32D1 (n= 11) | 277 (117)
  EOT (n= 347) | 144 (101)
  120 days after EOT (n= 124) | 10.4 (20.0)

16. Secondary Outcome: Time to Deterioration (TTD) in Patient-Reported Lung Cancer Symptoms, Using the European Organization for Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire (QLQ) Lung Cancer Supplemental Module 13 (LC13)
Description: TTD in patient-reported lung cancer symptoms (pain in chest or in arm/shoulder, dyspnea, or cough) was a composite endpoint defined as the time from randomization to the earliest time the participant's scale scores showed a 10 point or greater increase after baseline in any of the symptoms. A >/=10-point change in the score perceived by participants was considered as clinically significant. The QLQ-LC13 consisted of 1 multi-item scale and 9 single items that assessed the specific symptoms (dyspnea, cough, hemoptysis, and site specific pain), side effects (sore mouth, dysphagia, neuropathy, and alopecia), and pain medication use of lung cancer participants receiving chemotherapy. Scale score range: 0 to 100. Higher symptom score = greater degree of symptom severity.
Time Frame: Day 1 of each treatment Cycle up to EOT (up to approximately 2.25 years) (1 Cycle = 21 days)
Population: The PP-ITT analysis set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Months
  Pain in Chest | 8.3 [4.6 to 12.5] | 18.0 [11.0 to NA] — Data not reported because the upper limit of CI was not estimable due to higher number of censored participants.
  Cough | 5.6 [4.0 to 12.8] | 5.5 [4.2 to 7.9]
  Dyspnea | 2.1 [1.6 to 2.3] | 1.8 [1.5 to 2.3]
  Arm/Shoulder Pain | 6.2 [4.9 to 14.7] | 8.3 [5.8 to 12.8]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; Pain in Chest: Stratified analysis based on the strata of IC levels per IxRS, the number of prior chemotherapy regimens per IxRS, and histology per eCRF; Test type: Superiority or Other; p = 0.0111, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.55 to 0.93]
Statistical Analysis 2: Comparison: Docetaxel vs Atezolizumab; Cough: Unstratified Analysis; Test type: Superiority or Other; p = 0.6305, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.84 to 1.33]
Statistical Analysis 3: Comparison: Docetaxel vs Atezolizumab; Dyspnea: Unstratified Analysis; Test type: Superiority or Other; p = 0.7406, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.81 to 1.16]
Statistical Analysis 4: Comparison: Docetaxel vs Atezolizumab; Arm/Shoulder Pain; Test type: Superiority or Other; p = 0.5221, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.73 to 1.17]

17. Secondary Outcome: EORTC QLQ Core 30 (C30) Questionnaire Score: Single Items
Description: EORTC QLQ-C30 included global health status (GHS)/quality of life (QOL), functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Most questions from QLQ-C30 were a 4-point scale (1/Not at All to 4/Very Much), except Items 29-30, which comprise GHS scale and were a 7-point scale (1/Very Poor to 7/Excellent). For this instrument, GHS/QOL and functional scales were linearly transformed so each score ranged 0-100, where lower scores indicate poorer functioning (e.g., worsening) and higher scores indicate better functioning (e.g., improvement). Symptom scales/items were also linearly transformed so each score ranged 0-100, where higher scores indicate worse symptoms (e.g., more severe/worsened) and lower scores indicate less symptoms (e.g., less severe/improvement).
Time Frame: Day 1 of each treatment Cycle up to EOT (up to approximately 2.25 years); 6 week following PD ( Pro Week 6 Pd) (up to approximately 2.25 years); survival follow-up-1 (up to approximately 2.25 years) (1 Cycle= 21 days)
Population: The PP-ITT analysis set. Here, 'n' signifies those participants evaluated for this measure at specific time point for each group respectively. All 850 participants contributed to the endpoint but not all completed evaluation of every timepoint. Convention 'CxDx' refers to cycle number and day number.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Appetite Loss: Baseline (n= 390, 413) | 26.58 (31.57) | 22.92 (29.41)
  Appetite Loss: Cycle (C) 2 Day (D) 1(n= 342, 368) | 27.49 (30.39) | 26.99 (31.16)
  Appetite Loss: C3D1(n= 256, 304) | 21.35 (28.84) | 21.16 (28.94)
  Appetite Loss: C4D1(n= 224, 279) | 18.75 (25.36) | 18.40 (26.60)
  Appetite Loss: C5D1(n= 166, 238) | 18.88 (23.89) | 16.67 (27.52)
  Appetite Loss: C6D1(n= 151, 224) | 18.98 (25.68) | 14.88 (25.39)
  Appetite Loss: C7D1(n= 88, 190) | 15.91 (24.75) | 12.46 (23.06)
  Appetite Loss: C8D1(n= 72, 170) | 13.89 (22.20) | 12.94 (23.27)
  Appetite Loss: C9D1(n= 50, 153) | 8.00 (18.52) | 11.33 (22.35)
  Appetite Loss: C10D1(n= 47, 146) | 7.80 (15.87) | 12.33 (21.45)
  Appetite Loss: C11D1(n= 37, 134) | 11.71 (23.85) | 11.44 (22.43)
  Appetite Loss: C12D1(n= 30, 132) | 11.11 (20.22) | 8.84 (18.81)
  Appetite Loss: C13D1(n= 19, 123) | 10.53 (15.92) | 8.40 (15.74)
  Appetite Loss: C14D1(n= 18, 120) | 7.41 (14.26) | 10.00 (17.61)
  Appetite Loss: C15D1(n= 16, 113) | 6.25 (13.44) | 12.39 (22.80)
  Appetite Loss: C16D1(n= 13, 109) | 7.69 (14.62) | 10.09 (19.51)
  Appetite Loss: C17D1(n= 11, 98) | 6.06 (13.48) | 7.82 (18.41)
  Appetite Loss: C18D1(n= 10, 91) | 6.67 (14.05) | 8.06 (18.15)
  Appetite Loss: C19D1(n= 9, 84) | 7.41 (14.70) | 9.13 (18.18)
  Appetite Loss: C20D1(n= 9, 80) | 11.11 (23.57) | 9.58 (21.34)
  Appetite Loss: C21D1(n= 9, 75) | 3.70 (11.11) | 12.44 (26.15)
  Appetite Loss: C22D1(n= 8, 69) | 8.33 (15.43) | 6.76 (16.74)
  Appetite Loss: C23D1(n= 8, 66) | 8.33 (15.43) | 7.58 (17.34)
  Appetite Loss: C24D1(n= 5, 64) | 13.33 (18.26) | 8.33 (15.71)
  Appetite Loss: C25D1(n= 3, 60) | 0.00 (0.00) | 6.11 (13.01)
  Appetite Loss: C26D1(n= 3, 55) | 22.22 (19.24) | 5.45 (12.45)
  Appetite Loss: C27D1(n= 3, 52) | 0.00 (0.00) | 9.62 (19.06)
  Appetite Loss: C28D1(n= 1, 49) | 0.00 (NA) — Data not reported because standard deviation (SD) was non-estimable since only 1 participant was evaluated for this category. | 7.48 (15.61)
  Appetite Loss: C29D1(n= 2, 40) | 33.33 (47.14) | 9.17 (16.86)
  Appetite Loss: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 1.08 (5.99)
  Appetite Loss: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.94 (13.83)
  Appetite Loss: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 7.58 (22.84)
  Appetite Loss: C33D1(n= 0,16) | NA (NA) — Data not reported because no participant was evaluated for this category | 8.33 (25.82)
  Appetite Loss: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.76 (17.82)
  Appetite Loss: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 8.33 (20.72)
  Appetite Loss: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.78)
  Appetite Loss: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.67 (14.91)
  Appetite Loss: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Appetite Loss: End of treatment (EOT)(n= 265, 246) | 29.81 (31.85) | 31.98 (33.51)
  Appetite Loss: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Appetite Loss: Survival Follow-up (FU) 1 (n= 2, 1) | 50.00 (70.71) | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Constipation: Baseline (n= 388, 410) | 19.93 (27.39) | 16.50 (26.81)
  Constipation: C2D1(n= 339, 363) | 19.47 (26.42) | 18.09 (26.92)
  Constipation: C3D1(n= 255, 304) | 19.74 (26.91) | 15.13 (23.71)
  Constipation: C4D1(n= 224, 277) | 17.86 (23.38) | 14.56 (23.58)
  Constipation: C5D1(n= 166, 236) | 13.05 (21.33) | 12.15 (21.16)
  Constipation: C6D1(n= 151, 225) | 14.35 (23.89) | 12.89 (22.42)
  Constipation: C7D1(n= 87, 188) | 13.41 (20.62) | 11.52 (21.04)
  Constipation: C8D1(n= 72, 171) | 8.33 (15.57) | 12.28 (21.36)
  Constipation: C9D1(n= 50, 153) | 9.33 (19.10) | 10.68 (17.79)
  Constipation: C10D1(n= 47, 146) | 9.22 (17.99) | 9.82 (17.58)
  Constipation: C11D1(n= 37, 134) | 5.41 (12.46) | 9.95 (17.83)
  Constipation: C12D1(n= 30, 132) | 11.11 (20.22) | 10.86 (18.65)
  Constipation: C13D1(n= 19, 124) | 5.26 (12.49) | 8.60 (15.83)
  Constipation: C14D1(n= 17, 121) | 15.69 (23.91) | 9.09 (16.67)
  Constipation: C15D1(n= 15, 113) | 2.22 (8.61) | 10.03 (17.75)
  Constipation: C16D1(n= 13, 109) | 20.51 (32.03) | 9.79 (18.87)
  Constipation: C17D1(n= 11, 98) | 12.12 (22.47) | 9.86 (19.27)
  Constipation: C18D1(n= 10, 92) | 6.67 (14.05) | 9.06 (17.89)
  Constipation: C19D1(n= 9, 83) | 7.41 (14.70) | 9.64 (18.43)
  Constipation: C20D1(n=9, 80) | 14.81 (33.79) | 12.50 (23.35)
  Constipation: C21D1(n= 9, 75) | 7.41 (14.70) | 14.22 (25.22)
  Constipation: C22D1(n= 8, 69) | 12.50 (24.80) | 11.59 (21.26)
  Constipation: C23D1(n= 8, 66) | 4.17 (11.78) | 10.10 (20.23)
  Constipation: C24D1(n=5, 65) | 20.00 (29.81) | 9.74 (17.40)
  Constipation: C25D1(n= 3, 60) | 0.00 (0.00) | 11.11 (19.08)
  Constipation: C26D1(n= 2, 55) | 0.00 (0.00) | 12.12 (20.65)
  Constipation: C27D1(n= 3, 52) | 0.00 (0.00) | 13.46 (20.09)
  Constipation: C28D1(n= 1, 48) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 11.81 (22.27)
  Constipation: C29D1(n= 2, 40) | 50.00 (70.71) | 15.83 (23.86)
  Constipation: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 8.60 (19.18)
  Constipation: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 9.72 (20.80)
  Constipation: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.06 (13.16)
  Constipation: C33D1(n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.39)
  Constipation: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 7.14 (14.19)
  Constipation: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 5.56 (12.97)
  Constipation: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.78)
  Constipation: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Constipation: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Constipation: EOT (n= 265, 246) | 19.12 (27.28) | 19.78 (28.36)
  Constipation: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Constipation: Survival FU-1 (n= 2,1) | 33.33 (47.14) | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Diarrhea: Baseline (n= 388, 411) | 5.84 (13.77) | 7.22 (17.86)
  Diarrhea: C2D1(n= 339, 361) | 11.21 (20.65) | 7.29 (17.72)
  Diarrhea: C3D1(n= 255, 304) | 10.07 (18.68) | 6.14 (15.75)
  Diarrhea: C4D1(n= 223, 280) | 8.22 (16.35) | 6.67 (17.71)
  Diarrhea: C5D1(n= 166, 238) | 8.43 (17.48) | 6.58 (16.16)
  Diarrhea: C6D1(n= 151, 222) | 7.51 (14.99) | 6.31 (14.88)
  Diarrhea: C7D1(n= 87, 189) | 10.34 (17.10) | 7.94 (17.24)
  Diarrhea: C8D1(n= 72, 171) | 7.41 (15.03) | 8.77 (17.56)
  Diarrhea: C9D1(n= 50, 153) | 11.33 (17.31) | 7.63 (16.44)
  Diarrhea: C10D1(n= 47, 146) | 7.80 (14.27) | 5.48 (15.67)
  Diarrhea: C11D1(n= 36, 134) | 8.33 (14.64) | 4.98 (14.46)
  Diarrhea: C12D1(n= 30, 132) | 10.00 (17.83) | 6.31 (16.54)
  Diarrhea: C13D1(n= 18, 124) | 11.11 (16.17) | 5.65 (14.55)
  Diarrhea: C14D1(n= 17, 121) | 3.92 (11.07) | 9.92 (19.07)
  Diarrhea: C15D1(n= 15, 113) | 8.89 (15.26) | 7.96 (17.97)
  Diarrhea: C16D1(n= 12, 108) | 13.89 (17.16) | 6.48 (14.02)
  Diarrhea: C17D1(n= 11, 98) | 9.09 (15.57) | 7.82 (16.44)
  Diarrhea: C18D1(n= 10, 92) | 13.33 (17.21) | 8.70 (17.73)
  Diarrhea: C19D1(n= 9, 84) | 14.81 (17.57) | 7.94 (18.38)
  Diarrhea: C20D1(n= 9, 80) | 7.41 (14.70) | 6.67 (14.43)
  Diarrhea: C21D1(n= 9, 75) | 18.52 (17.57) | 11.11 (18.45)
  Diarrhea: C22D1(n= 8, 68) | 16.67 (25.20) | 7.84 (16.41)
  Diarrhea: C23D1(n= 8, 66) | 8.33 (15.43) | 6.06 (16.44)
  Diarrhea: C24D1(n= 5, 64) | 6.67 (14.91) | 6.25 (16.67)
  Diarrhea: C25D1(n= 3, 60) | 0.00 (0.00) | 6.11 (14.38)
  Diarrhea: C26D1(n= 3, 55) | 11.11 (19.24) | 10.30 (21.15)
  Diarrhea: C27D1(n= 3, 52) | 11.11 (19.24) | 5.77 (15.79)
  Diarrhea: C28D1(n= 1, 48) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 4.86 (13.73)
  Diarrhea: C29D1(n= 2, 40) | 50.00 (70.71) | 9.17 (18.47)
  Diarrhea: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 7.53 (16.58)
  Diarrhea: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.94 (16.97)
  Diarrhea: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 12.12 (16.41)
  Diarrhea: C33D1(n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 8.33 (14.91)
  Diarrhea: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.76 (12.10)
  Diarrhea: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 5.56 (12.97)
  Diarrhea: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.78)
  Diarrhea: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.67 (14.91)
  Diarrhea: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Diarrhea: EOT(n= 265, 246) | 10.57 (19.18) | 9.35 (20.39)
  Diarrhea: Pro Week 6 Pd(n= 0, 1) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Diarrhea: Survival FU-1 (n= 2, 1) | 33.33 (47.14) | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Financial Difficulties: Baseline (n=387, 411) | 20.76 (27.61) | 18.09 (28.32)
  Financial Difficulties: C2D1 (n=336, 362) | 18.45 (26.20) | 15.93 (26.28)
  Financial Difficulties: C3D1 (n=253, 305) | 16.86 (24.24) | 15.63 (25.79)
  Financial Difficulties: C4D1 (n=219, 280) | 16.74 (23.97) | 15.12 (24.72)
  Financial Difficulties: C5D1 (n=165, 238) | 16.57 (24.03) | 15.13 (25.71)
  Financial Difficulties: C6D1 (n=149, 224) | 15.66 (24.06) | 16.67 (26.41)
  Financial Difficulties: C7D1 (n=86, 189) | 16.28 (24.92) | 17.46 (27.41)
  Financial Difficulties: C8D1 (n=71, 170) | 13.15 (21.44) | 18.82 (27.59)
  Financial Difficulties: C9D1 (n=49, 152) | 16.33 (28.16) | 17.54 (27.38)
  Financial Difficulties: C10D1 (n=46, 146) | 14.49 (23.99) | 17.81 (29.08)
  Financial Difficulties: C11D1 (n=36, 134) | 9.26 (21.98) | 19.65 (30.10)
  Financial Difficulties: C12D1 (n=30, 132) | 12.22 (23.95) | 18.43 (28.92)
  Financial Difficulties: C13D1 (n=18, 122) | 12.96 (25.92) | 18.31 (29.10)
  Financial Difficulties: C14D1 (n=17, 121) | 15.69 (26.66) | 18.46 (29.17)
  Financial Difficulties: C15D1 (n=15, 113) | 6.67 (18.69) | 18.29 (28.86)
  Financial Difficulties: C16D1 (n=12, 109) | 13.89 (30.01) | 18.65 (29.20)
  Financial Difficulties: C17D1 (n=11, 98) | 15.15 (22.92) | 18.37 (27.55)
  Financial Difficulties: C18D1 (n=10, 92) | 10.00 (22.50) | 19.57 (28.45)
  Financial Difficulties: C19D1 (n=9, 84) | 3.70 (11.11) | 19.05 (28.94)
  Financial Difficulties: C20D1 (n=9, 80) | 11.11 (33.33) | 18.75 (27.99)
  Financial Difficulties: C21D1 (n=9, 75) | 11.11 (33.33) | 23.11 (30.99)
  Financial Difficulties: C22D1 (n=8, 68) | 12.50 (35.36) | 18.63 (28.44)
  Financial Difficulties: C23D1 (n=7, 66) | 9.52 (25.20) | 21.72 (30.66)
  Financial Difficulties: C24D1 (n=5, 64) | 13.33 (29.81) | 20.83 (29.99)
  Financial Difficulties: C25D1 (n=3, 60) | 0.00 (0.00) | 21.67 (31.19)
  Financial Difficulties: C26D1 (n=3, 55) | 0.00 (0.00) | 20.00 (30.50)
  Financial Difficulties: C27D1 (n=3, 52) | 0.00 (0.00) | 17.31 (28.38)
  Financial Difficulties: C28D1 (n=1, 48) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 18.06 (26.59)
  Financial Difficulties: C29D1 (n=2, 40) | 50.00 (70.71) | 19.17 (28.13)
  Financial Difficulties: C30D1 (n=1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 17.20 (25.63)
  Financial Difficulties: C31D1(n=0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 20.83 (25.66)
  Financial Difficulties: C32D1(n=0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 21.21 (26.32)
  Financial Difficulties: C33D1(n=0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 22.92 (29.11)
  Financial Difficulties: C34D1(n=0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 26.19 (35.03)
  Financial Difficulties: C35D1(n=0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 27.78 (37.15)
  Financial Difficulties: C36D1(n=0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 8.33 (15.43)
  Financial Difficulties: C37D1(n=0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 26.67 (43.46)
  Financial Difficulties: C38D1(n=0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 16.67 (23.57)
  Financial Difficulties: EOT(n=263, 245) | 21.80 (29.23) | 19.46 (28.75)
  Financial Difficulties: Pro Week 6 Pd (n=0, 1) | NA (NA) — Data not reported because no participant was evaluated for this category | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Financial Difficulties:Survival FU-1 (n=2,24) | 83.33 (23.57) | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Insomnia: Baseline (n= 388, 413) | 28.87 (30.55) | 26.15 (28.72)
  Insomnia: C2D1(n= 340, 367) | 27.55 (30.87) | 26.52 (28.61)
  Insomnia: C3D1(n= 253, 304) | 25.69 (29.15) | 24.89 (27.32)
  Insomnia: C4D1(n= 222, 279) | 21.32 (26.07) | 23.66 (26.48)
  Insomnia: C5D1(n= 166, 237) | 21.49 (25.43) | 25.88 (29.84)
  Insomnia: C6D1(n= 150, 225) | 22.00 (26.71) | 23.41 (27.73)
  Insomnia: C7D1(n= 87, 189) | 21.07 (25.47) | 23.99 (26.65)
  Insomnia: C8D1(n= 70, 169) | 15.24 (23.87) | 23.87 (26.27)
  Insomnia: C9D1(n= 49, 153) | 16.33 (26.46) | 22.88 (27.16)
  Insomnia: C10D1(n= 46, 144) | 13.77 (19.34) | 21.53 (26.87)
  Insomnia: C11D1(n= 36, 133) | 9.26 (18.87) | 20.55 (27.44)
  Insomnia: C12D1(n= 29, 132) | 16.09 (30.37) | 21.46 (24.41)
  Insomnia: C13D1(n= 17, 124) | 17.65 (29.15) | 23.39 (28.51)
  Insomnia: C14D1(n= 17, 121) | 25.49 (27.71) | 23.69 (26.33)
  Insomnia: C15D1(n= 15, 113) | 22.22 (29.99) | 21.53 (28.84)
  Insomnia: C16D1(n= 13, 108) | 20.51 (25.60) | 21.60 (31.01)
  Insomnia: C17D1(n= 11, 98) | 21.21 (26.97) | 20.07 (28.21)
  Insomnia: C18D1(n= 10, 92) | 20.00 (32.20) | 21.38 (27.77)
  Insomnia: C19D1(n= 9, 83) | 18.52 (24.22) | 22.49 (28.09)
  Insomnia: C20D1(n= 9, 80) | 18.52 (33.79) | 20.83 (29.71)
  Insomnia: C21D1(n= 9, 75) | 22.22 (33.33) | 20.89 (29.90)
  Insomnia: C22D1(n= 8, 69) | 16.67 (35.63) | 18.84 (26.49)
  Insomnia: C23D1(n= 8, 66) | 20.83 (35.36) | 19.70 (28.03)
  Insomnia: C24D1(n= 5, 64) | 26.67 (27.89) | 19.79 (25.00)
  Insomnia: C25D1(n= 3, 60) | 11.11 (19.24) | 18.89 (23.26)
  Insomnia: C26D1(n= 3, 55) | 11.11 (19.24) | 21.21 (27.49)
  Insomnia: C27D1(n= 3, 52) | 11.11 (19.24) | 19.23 (28.27)
  Insomnia: C28D1(n= 1, 49) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 21.09 (27.80)
  Insomnia: C29D1(n= 2, 40) | 33.33 (47.14) | 21.67 (26.74)
  Insomnia: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 20.43 (28.12)
  Insomnia: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 20.83 (27.47)
  Insomnia: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 19.70 (26.55)
  Insomnia: C33D1(n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 20.83 (34.16)
  Insomnia: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 23.81 (24.21)
  Insomnia: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 25.00 (28.87)
  Insomnia: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 25.00 (23.57)
  Insomnia: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 33.33 (23.57)
  Insomnia: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 16.67 (23.57)
  Insomnia: EOT(n= 264, 246) | 28.91 (30.65) | 29.95 (30.30)
  Insomnia: Pro Week Pd(n= 0, 1) | NA (NA) — Data not reported because no participant was evaluated for this category | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Insomnia: Survival FU-1 (n= 2, 1) | 50.00 (70.71) | 100.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Dyspnea: C1D1 (n= 389, 412) | 33.50 (31.11) | 32.04 (28.73)
  Dyspnea: C2D1 (n= 341, 368) | 32.55 (29.03) | 31.88 (29.70)
  Dyspnea: C3D1 (n= 255, 302) | 29.93 (27.54) | 27.15 (26.73)
  Dyspnea: C4D1 (n= 389, 277) | 28.38 (24.37) | 28.28 (27.48)
  Dyspnea: C5D1 (n= 222, 236) | 29.52 (24.46) | 27.82 (27.03)
  Dyspnea: C6D1 (n= 166, 222) | 30.02 (26.32) | 26.88 (25.63)
  Dyspnea: C7D1 (n= 151, 188) | 27.13 (25.31) | 25.53 (25.99)
  Dyspnea: C8D1 (n= 86, 169) | 28.70 (29.76) | 26.43 (26.70)
  Dyspnea: C9D1 (n= 72, 152) | 26.67 (28.57) | 24.12 (24.92)
  Dyspnea: C10D1 (n= 50, 146) | 27.66 (28.93) | 23.52 (23.54)
  Dyspnea: C11D1 (n= 47, 134) | 25.23 (30.84) | 22.89 (25.00)
  Dyspnea: C12D1 (n= 37, 132) | 26.67 (26.84) | 22.73 (25.83)
  Dyspnea: C13D1 (n= 30, 123) | 19.30 (23.08) | 25.47 (26.68)
  Dyspnea: C14D1 (n= 19, 119) | 20.37 (25.92) | 21.85 (25.47)
  Dyspnea: C15D1 (n= 16, 113) | 16.67 (17.21) | 22.71 (24.51)
  Dyspnea: C16D1 (n= 13, 109) | 20.51 (16.88) | 21.71 (25.00)
  Dyspnea: C17D1 (n= 11, 98) | 15.15 (17.41) | 21.43 (23.57)
  Dyspnea: C18D1 (n= 10, 92) | 20.00 (17.21) | 22.83 (25.64)
  Dyspnea: C19D1 (n= 9, 84) | 11.11 (16.67) | 23.41 (23.59)
  Dyspnea: C20D1 (n= 9, 80) | 18.52 (17.57) | 21.67 (24.36)
  Dyspnea: C21D1 (n= 9, 75) | 18.52 (17.57) | 19.11 (20.63)
  Dyspnea: C22D1 (n= 8, 68) | 20.83 (35.36) | 20.59 (23.06)
  Dyspnea: C23D1 (n= 8, 65) | 12.50 (17.25) | 18.46 (21.27)
  Dyspnea: C24D1 (n= 5, 64) | 6.67 (14.91) | 19.79 (24.28)
  Dyspnea: C25D1 (n= 3, 60) | 11.11 (19.24) | 20.00 (22.30)
  Dyspnea: C26D1 (n= 3, 55) | 0.00 (0.00) | 20.00 (24.51)
  Dyspnea: C27D1 (n= 3, 52) | 0.00 (0.00) | 16.03 (19.23)
  Dyspnea: C28D1 (n= 1, 49) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 17.01 (20.55)
  Dyspnea: C29D1 (n= 2, 40) | 33.33 (47.14) | 15.00 (21.28)
  Dyspnea: C30D1 (n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 16.13 (18.99)
  Dyspnea: C31D1 (n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 22.22 (23.40)
  Dyspnea: C32D1 (n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 22.73 (21.54)
  Dyspnea: C33D1 (n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 25.00 (31.03)
  Dyspnea: C34D1 (n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 26.19 (26.73)
  Dyspnea: C35D1 (n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 25.00 (25.13)
  Dyspnea: C36D1 (n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 20.83 (17.25)
  Dyspnea: C37D1 (n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 26.67 (14.91)
  Dyspnea: C38D1 (n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 33.33 (0.00)
  Dyspnea: EOT(n= 266, 247) | 38.72 (30.51) | 39.41 (32.57)
  Dyspnea: Pro Week 6 Pd (n= 0, 1) | NA (NA) — Data not reported because no participant was evaluated for this category | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Dyspnea: Survival Follow-Up 1 (n= 2, 1) | 33.33 (47.14) | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

18. Secondary Outcome: EORTC QLQ-C30 Questionnaire Score: Functional Subscales
Description: EORTC QLQ-C30 included GHS/QOL, functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Most questions from QLQ-C30 were a 4-point scale (1/Not at All to 4/Very Much), except Items 29-30, which comprise GHS scale and were a 7-point scale (1/Very Poor to 7/Excellent). For this instrument, GHS/QOL and functional scales were linearly transformed so each score ranged 0-100, where lower scores indicate poorer functioning (e.g., worsening) and higher scores indicate better functioning (e.g., improvement). Symptom scales/items were also linearly transformed so each score ranged 0-100, where higher scores indicate worse symptoms (e.g., more severe/worsened) and lower scores indicate less symptoms (e.g., less severe/improvement).
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Cognitive: Baseline (n= 390, 411) | 83.38 (20.68) | 85.16 (19.16)
  Cognitive: C2D1 (n= 341, 363) | 83.38 (21.64) | 84.94 (19.30)
  Cognitive: C3D1(n= 256, 305) | 84.05 (19.82) | 86.28 (17.32)
  Cognitive: C4D1(n= 224, 281) | 84.82 (19.27) | 85.35 (19.87)
  Cognitive: C5D1(n= 166, 238) | 86.04 (17.24) | 84.38 (19.73)
  Cognitive: C6D1(n= 151, 224) | 86.09 (18.20) | 84.45 (20.27)
  Cognitive: C7D1(n= 87, 189) | 87.55 (16.32) | 84.74 (18.93)
  Cognitive: C8D1(n= 72, 171) | 89.58 (13.83) | 85.58 (18.87)
  Cognitive: C9D1(n= 50, 153) | 90.00 (14.29) | 85.95 (18.65)
  Cognitive: C10D1(n= 47, 146) | 91.13 (11.96) | 86.53 (19.31)
  Cognitive: C11D1(n= 36, 134) | 92.59 (10.87) | 85.95 (19.91)
  Cognitive: C12D1(n= 30, 132) | 91.11 (12.17) | 84.22 (20.52)
  Cognitive: C13D1(n= 18, 124) | 90.74 (11.75) | 84.27 (21.50)
  Cognitive: C14D1(n= 17, 121) | 92.16 (11.96) | 85.67 (18.30)
  Cognitive: C15D1(n= 15, 113) | 93.33 (10.54) | 85.10 (19.08)
  Cognitive: C16D1(n= 12, 109) | 97.22 (6.49) | 85.32 (21.12)
  Cognitive: C17D1(n= 11, 98) | 96.97 (6.74) | 85.37 (20.48)
  Cognitive: C18D1(n= 10, 92) | 91.67 (11.79) | 82.97 (20.52)
  Cognitive: C19D1(n= 9, 84) | 92.59 (12.11) | 83.53 (20.12)
  Cognitive: C20D1(n= 9, 80) | 90.74 (14.70) | 82.29 (22.87)
  Cognitive: C21D1(n= 9, 75) | 87.04 (23.24) | 83.78 (20.32)
  Cognitive: C22D1(n= 8, 68) | 89.58 (12.40) | 84.56 (21.03)
  Cognitive: C23D1(n= 8, 66) | 95.83 (7.72) | 84.09 (20.55)
  Cognitive: C24D1(n= 5, 64) | 83.33 (23.57) | 83.85 (23.56)
  Cognitive: C25D1(n= 3, 60) | 72.22 (25.46) | 83.61 (21.59)
  Cognitive: C26D1(n= 3, 55) | 77.78 (19.24) | 82.73 (21.51)
  Cognitive: C27D1(n= 3, 52) | 88.89 (19.24) | 85.26 (20.25)
  Cognitive: C28D1(n= 1, 48) | 100.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 85.07 (20.98)
  Cognitive: C29D1(n= 2, 40) | 50.00 (70.71) | 83.75 (20.84)
  Cognitive: C30D1(n= 1, 31) | 100.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 86.02 (20.68)
  Cognitive: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 80.56 (21.23)
  Cognitive: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 82.58 (22.11)
  Cognitive: C33D1(n= 0,16) | NA (NA) — Data not reported because no participant was evaluated for this category | 77.08 (25.73)
  Cognitive: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 80.95 (24.33)
  Cognitive: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 76.39 (21.86)
  Cognitive: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 83.33 (15.43)
  Cognitive: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 83.33 (16.67)
  Cognitive: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 91.67 (11.79)
  Cognitive: EOT (n= 266, 246) | 78.82 (24.54) | 78.52 (22.50)
  Cognitive: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 83.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Cognitive: Survival FU 1 (n= 2, 1) | 50.00 (47.14) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Emotional: Baseline (n= 390, 411) | 75.83 (22.59) | 76.55 (21.77)
  Emotional: C2D1(n= 341, 363) | 78.06 (22.63) | 79.47 (20.72)
  Emotional: C3D1(n= 256, 305) | 79.70 (22.24) | 82.71 (17.45)
  Emotional: C4D1(n= 224, 280) | 81.67 (20.36) | 83.69 (17.70)
  Emotional: C5D1(n= 166, 238) | 80.52 (20.24) | 81.99 (19.22)
  Emotional: C6D1(n= 151, 224) | 81.73 (20.50) | 82.70 (19.91)
  Emotional: C7D1(n= 87, 189) | 81.42 (22.00) | 83.77 (17.71)
  Emotional: C8D1(n= 72, 171) | 84.38 (18.66) | 83.63 (19.40)
  Emotional: C9D1(n= 50, 153) | 86.00 (17.93) | 85.62 (18.72)
  Emotional: C10D1(n= 47, 146) | 84.93 (17.69) | 84.13 (19.74)
  Emotional: C11D1(n= 36, 134) | 89.12 (15.15) | 84.16 (18.14)
  Emotional: C12D1(n= 30, 132) | 86.94 (14.79) | 84.34 (20.10)
  Emotional: C13D1(n= 18, 123) | 89.35 (14.52) | 84.35 (19.75)
  Emotional: C14D1(n= 17, 121) | 86.27 (15.57) | 84.25 (19.11)
  Emotional: C15D1(n= 15, 113) | 90.00 (14.16) | 83.87 (20.04)
  Emotional: C16D1(n= 12, 109) | 88.89 (16.02) | 82.11 (22.59)
  Emotional: C17D1(n= 11, 98) | 88.64 (17.59) | 83.25 (19.50)
  Emotional: C18D1(n= 10, 92) | 87.50 (19.35) | 82.52 (21.11)
  Emotional: C19D1(n= 9, 84) | 87.96 (19.14) | 81.42 (20.55)
  Emotional: C20D1(n=9, 80) | 76.85 (34.30) | 83.19 (18.90)
  Emotional: C21D1(n= 9, 75) | 83.33 (26.68) | 84.19 (17.58)
  Emotional: C22D1(n= 8, 68) | 76.74 (32.60) | 86.03 (16.44)
  Emotional: C23D1(n= 8, 66) | 89.58 (15.91) | 87.00 (17.55)
  Emotional: C24D1(n=5, 65) | 78.33 (33.12) | 83.72 (19.18)
  Emotional: C25D1(n= 3, 60) | 100.00 (0.00) | 83.66 (18.77)
  Emotional: C26D1(n= 3, 55) | 86.11 (12.73) | 85.15 (19.69)
  Emotional: C27D1(n= 3, 52) | 100.00 (0.00) | 86.38 (18.38)
  Emotional: C28D1(n= 1, 48) | 100.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 86.92 (17.51)
  Emotional: C29D1(n= 2, 40) | 50.00 (70.71) | 87.50 (16.45)
  Emotional: C30D1(n= 1, 31) | 100.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 89.79 (15.62)
  Emotional: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 85.76 (18.30)
  Emotional: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 82.95 (20.81)
  Emotional: C33D1(n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 81.25 (25.37)
  Emotional: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 82.14 (25.29)
  Emotional: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 83.33 (21.61)
  Emotional: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 95.83 (11.78)
  Emotional: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 90.00 (14.91)
  Emotional: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 83.33 (23.57)
  Emotional: EOT (n= 265, 246) | 73.78 (26.29) | 73.92 (23.74)
  Emotional: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Emotional: Survival FU-1 (n= 2,1) | 25.00 (35.36) | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Physical: Baseline (n= 390, 413) | 73.27 (22.58) | 74.46 (20.66)
  Physical: C2D1(n= 343, 369) | 72.64 (22.00) | 71.70 (22.49)
  Physical: C3D1(n= 255, 304) | 74.98 (21.60) | 76.19 (19.48)
  Physical: C4D1(n= 224, 277) | 75.72 (19.05) | 76.79 (19.95)
  Physical: C5D1(n= 167, 238) | 77.30 (19.00) | 77.79 (19.89)
  Physical: C6D1(n= 151, 225) | 74.77 (19.26) | 78.93 (18.76)
  Physical: C7D1(n= 88, 189) | 77.61 (18.08) | 79.20 (18.42)
  Physical: C8D1(n= 71, 170) | 78.45 (17.72) | 78.87 (18.91)
  Physical: C9D1(n= 50, 153) | 79.07 (20.43) | 79.46 (18.75)
  Physical: C10D1(n= 47, 146) | 79.29 (19.96) | 79.41 (18.85)
  Physical: C11D1(n= 37, 134) | 81.44 (20.85) | 79.09 (20.50)
  Physical: C12D1(n= 30, 132) | 82.22 (15.69) | 79.72 (18.84)
  Physical: C13D1(n= 19, 124) | 87.37 (9.66) | 80.48 (19.33)
  Physical: C14D1(n= 18, 121) | 85.56 (9.50) | 80.33 (17.55)
  Physical: C15D1(n= 16, 113) | 86.25 (8.24) | 79.88 (18.64)
  Physical: C16D1(n= 13, 109) | 85.13 (9.49) | 78.82 (21.32)
  Physical: C17D1(n= 11, 98) | 84.24 (12.03) | 78.57 (20.89)
  Physical: C18D1(n= 10, 92) | 82.67 (13.03) | 79.64 (19.92)
  Physical: C19D1(n= 9, 84) | 87.41 (10.77) | 78.97 (20.48)
  Physical: C20D1(n= 9, 80) | 81.48 (18.19) | 79.19 (20.26)
  Physical: C21D1(n= 9, 75) | 87.41 (11.28) | 78.67 (20.68)
  Physical: C22D1(n= 8, 69) | 82.50 (19.82) | 82.51 (16.92)
  Physical: C23D1(n= 8, 66) | 85.00 (13.21) | 80.81 (17.56)
  Physical: C24D1(n= 5, 64) | 80.00 (18.26) | 81.41 (17.69)
  Physical: C25D1(n= 3, 60) | 82.22 (16.78) | 83.22 (16.67)
  Physical: C26D1(n= 3, 55) | 75.56 (3.85) | 80.12 (17.43)
  Physical: C27D1(n= 2, 52) | 76.67 (4.71) | 81.89 (16.90)
  Physical: C28D1(n= 2, 49) | 65.00 (21.21) | 84.15 (14.41)
  Physical: C29D1(n= 2, 40) | 56.67 (33.00) | 83.00 (14.87)
  Physical: C30D1(n= 1, 31) | 80.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 83.01 (15.67)
  Physical: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 78.61 (17.25)
  Physical: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 75.15 (18.42)
  Physical: C33D1(n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 77.92 (17.84)
  Physical: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 75.24 (19.47)
  Physical: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 73.89 (20.78)
  Physical: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 83.33 (17.46)
  Physical: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 74.67 (14.45)
  Physical: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 86.67 (0.00)
  Physical: EOT(n= 267, 246) | 63.59 (24.57) | 64.78 (26.47)
  Physical: Pro Week 6 Pd(n= 0, 1) | NA (NA) — Data not reported because no participant was evaluated for this category | 46.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Physical: Survival FU-1 (n= 2, 1) | 36.67 (51.85) | 46.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Role: Baseline (n=388, 413) | 70.92 (30.68) | 73.61 (29.13)
  Role: C2D1 (n=339, 369) | 69.91 (29.89) | 68.29 (31.50)
  Role: C3D1 (n=256, 304) | 74.61 (27.21) | 75.27 (27.28)
  Role: C4D1 (n=224, 279) | 73.36 (26.22) | 76.70 (25.27)
  Role: C5D1 (n=167, 238) | 74.35 (25.00) | 76.05 (26.97)
  Role: C6D1 (n=151, 225) | 73.62 (26.62) | 77.70 (26.78)
  Role: C7D1 (n=88, 190) | 77.27 (23.19) | 79.04 (24.97)
  Role: C8D1 (n=72, 170) | 73.61 (26.50) | 77.35 (25.22)
  Role: C9D1 (n=50, 153) | 77.67 (24.42) | 79.30 (25.36)
  Role: C10D1 (n=47, 145) | 78.72 (27.74) | 81.38 (24.34)
  Role: C11D1 (n=37, 134) | 80.63 (24.69) | 78.61 (27.01)
  Role: C12D1 (n=30, 132) | 81.11 (22.20) | 79.80 (25.97)
  Role: C13D1 (n=19, 124) | 84.21 (18.82) | 79.44 (26.55)
  Role: C14D1 (n=18, 121) | 78.70 (21.24) | 79.48 (24.98)
  Role: C15D1 (n=16, 113) | 83.33 (14.91) | 79.20 (25.05)
  Role: C16D1 (n=13, 109) | 85.90 (19.06) | 76.45 (27.89)
  Role: C17D1 (n=11, 98) | 80.30 (20.84) | 76.02 (29.22)
  Role: C18D1 (n=10, 92) | 80.00 (26.99) | 77.17 (27.59)
  Role: C19D1 (n=9, 84) | 85.19 (22.74) | 78.17 (28.46)
  Role: C20D1 (n=9, 80) | 79.63 (29.79) | 78.54 (26.01)
  Role: C21D1 (n=9, 75) | 85.19 (15.47) | 77.33 (28.29)
  Role: C22D1 (n=8, 69) | 79.17 (35.36) | 81.64 (26.68)
  Role: C23D1 (n=8, 66) | 85.42 (20.77) | 80.30 (26.13)
  Role: C24D1 (n=5, 65) | 70.00 (34.16) | 78.72 (26.92)
  Role: C25D1 (n=3, 60) | 77.78 (38.49) | 79.44 (27.34)
  Role: C26D1 (n=3, 55) | 83.33 (28.87) | 76.97 (27.31)
  Role: C27D1 (n=3, 52) | 88.89 (19.24) | 80.77 (26.89)
  Role: C28D1 (n=1, 49) | 100.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 82.99 (22.69)
  Role: C29D1 (n=2, 40) | 66.67 (47.14) | 83.33 (24.75)
  Role: C30D1 (n=1, 31) | 100.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 81.72 (24.10)
  Role: C31D1(n=0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 79.86 (25.53)
  Role: C32D1(n=0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 75.00 (27.58)
  Role: C33D1(n=0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 66.67 (34.43)
  Role: C34D1(n=0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 69.05 (33.88)
  Role: C35D1(n=0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 69.44 (32.44)
  Role: C36D1(n=0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 87.50 (17.25)
  Role: C37D1(n=0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 76.67 (22.36)
  Role: C38D1(n=0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 100.00 (0.00)
  Role: EOT(n=266, 246) | 58.52 (32.99) | 60.03 (33.25)
  Role: Pro Week 6 Pd (n=0, 1) | NA (NA) — Data not reported because no participant was evaluated for this category | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Role: Survival FU-1 (n=2,1) | 33.33 (47.14) | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Social: Baseline (n= 389, 411) | 74.16 (26.92) | 77.41 (26.13)
  Social: C2D1(n= 340, 363) | 74.51 (26.50) | 76.86 (26.25)
  Social: C3D1(n= 255, 305) | 78.37 (25.30) | 81.15 (23.70)
  Social: C4D1(n= 223, 280) | 79.60 (23.00) | 81.31 (24.15)
  Social: C5D1(n= 166, 238) | 79.32 (22.26) | 82.00 (24.39)
  Social: C6D1(n= 151, 224) | 78.15 (24.05) | 81.99 (23.80)
  Social: C7D1(n= 87, 189) | 80.65 (22.57) | 82.80 (22.54)
  Social: C8D1(n= 72, 171) | 81.94 (22.16) | 81.19 (23.95)
  Social: C9D1(n= 50, 153) | 82.00 (22.80) | 83.77 (22.29)
  Social: C10D1(n= 47, 146) | 81.21 (24.97) | 83.79 (22.99)
  Social: C11D1(n= 36, 134) | 82.41 (26.11) | 81.47 (25.42)
  Social: C12D1(n= 30, 132) | 86.67 (18.77) | 82.95 (24.58)
  Social: C13D1(n= 18, 124) | 89.81 (15.27) | 84.27 (22.82)
  Social: C14D1(n= 17, 121) | 86.27 (19.75) | 84.16 (22.55)
  Social: C15D1(n= 15, 113) | 93.33 (13.80) | 83.92 (22.26)
  Social: C16D1(n= 12, 109) | 84.72 (16.60) | 82.72 (24.73)
  Social: C17D1(n= 11, 98) | 87.88 (16.82) | 82.99 (23.57)
  Social: C18D1(n= 10, 92) | 86.67 (17.21) | 81.34 (24.06)
  Social: C19D1(n= 9, 84) | 88.89 (16.67) | 81.94 (25.90)
  Social: C20D1(n= 9, 80) | 81.48 (33.79) | 81.46 (24.73)
  Social: C21D1(n= 9, 75) | 85.19 (24.22) | 78.67 (27.88)
  Social: C22D1(n= 8, 68) | 85.42 (30.13) | 84.31 (25.41)
  Social: C23D1(n= 8, 66) | 91.67 (15.43) | 80.56 (26.24)
  Social: C24D1(n= 5, 65) | 80.00 (27.39) | 80.77 (25.38)
  Social: C25D1(n= 3, 60) | 77.78 (38.49) | 81.39 (27.80)
  Social: C26D1(n= 3, 55) | 77.78 (19.24) | 79.70 (27.53)
  Social: C27D1(n= 3, 52) | 88.89 (19.24) | 82.05 (25.32)
  Social: C28D1(n= 1, 48) | 100.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 84.03 (24.30)
  Social: C29D1(n= 2, 40) | 50.00 (70.71) | 82.92 (24.60)
  Social: C30D1(n= 1, 31) | 100.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 79.57 (27.79)
  Social: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 79.17 (26.12)
  Social: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 73.48 (30.71)
  Social: C33D1(n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 73.96 (32.19)
  Social: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 67.86 (34.88)
  Social: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 70.83 (31.88)
  Social: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 87.50 (17.25)
  Social: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 80.00 (18.26)
  Social: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 100.00 (0.00)
  Social: EOT(n= 264, 245) | 69.51 (30.65) | 70.00 (30.05)
  Social: Pro Week 6 Pd(n= 0, 1) | NA (NA) — Data not reported because no participant was evaluated for this category | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Social: Survival FU-1 (n= 2, 1) | 83.33 (23.57) | 16.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

19. Secondary Outcome: EORTC QLQ-C30 Questionnaire Score: GHS Scale
Description: as for outcome 18
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Global Health: Baseline (n= 387, 410) | 60.55 (22.25) | 61.24 (22.31)
  Global Health: C2D1(n= 339, 361) | 59.56 (22.15) | 58.93 (23.57)
  Global Health: C3D1(n= 255, 304) | 64.64 (18.66) | 64.61 (20.74)
  Global Health: C4D1(n= 222, 279) | 63.51 (20.67) | 65.11 (21.36)
  Global Health: C5D1(n= 166, 235) | 64.01 (18.37) | 66.35 (19.84)
  Global Health: C6D1(n= 151, 223) | 64.51 (19.59) | 65.73 (21.42)
  Global Health: C7D1(n= 87, 187) | 64.85 (18.13) | 66.93 (19.61)
  Global Health: C8D1(n= 72, 169) | 62.73 (20.22) | 67.36 (19.45)
  Global Health: C9D1(n= 50, 152) | 67.17 (18.93) | 68.09 (19.46)
  Global Health: C10D1(n= 47, 145) | 66.84 (18.67) | 69.37 (20.90)
  Global Health: C11D1(n= 36, 133) | 69.68 (17.15) | 68.17 (21.24)
  Global Health: C12D1(n= 30, 131) | 66.67 (18.05) | 68.32 (20.42)
  Global Health: C13D1(n= 18, 124) | 69.91 (14.33) | 67.74 (22.52)
  Global Health: C14D1(n= 17, 120) | 69.61 (14.71) | 67.01 (20.62)
  Global Health: C15D1(n= 15, 113) | 69.44 (17.16) | 68.66 (20.21)
  Global Health: C16D1(n= 12, 109) | 62.50 (15.69) | 67.97 (21.67)
  Global Health: C17D1(n= 10, 98) | 61.67 (19.72) | 68.62 (19.84)
  Global Health: C18D1(n= 10, 92) | 61.67 (21.23) | 68.57 (18.86)
  Global Health: C19D1(n= 9, 84) | 65.74 (21.43) | 68.25 (20.10)
  Global Health: C20D1(n= 9, 80) | 62.04 (26.72) | 68.12 (20.10)
  Global Health: C21D1(n= 9, 75) | 60.19 (29.98) | 66.56 (21.55)
  Global Health: C22D1(n= 8, 68) | 54.17 (24.80) | 73.28 (17.13)
  Global Health: C23D1(n= 8, 66) | 62.50 (19.42) | 70.45 (18.09)
  Global Health: C24D1(n= 5, 65) | 70.00 (27.39) | 69.36 (19.27)
  Global Health: C25D1(n= 3, 60) | 66.67 (28.87) | 69.03 (19.23)
  Global Health: C26D1(n= 3, 55) | 66.67 (28.87) | 68.64 (20.60)
  Global Health: C27D1(n= 3, 52) | 66.67 (28.87) | 68.91 (21.84)
  Global Health: C28D1(n= 2, 48) | 87.50 (17.68) | 71.87 (20.60)
  Global Health: C29D1(n= 2, 40) | 91.67 (11.79) | 72.71 (20.06)
  Global Health: C30D1(n= 1, 30) | 83.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 75.28 (18.63)
  Global Health: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 71.53 (21.13)
  Global Health: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 70.45 (20.21)
  Global Health: C33D1(n= 0,16) | NA (NA) — Data not reported because no participant was evaluated for this category | 67.19 (27.30)
  Global Health: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 68.45 (26.19)
  Global Health: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 69.44 (26.43)
  Global Health: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 80.21 (16.63)
  Global Health: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 76.67 (19.00)
  Global Health: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 91.67 (11.79)
  Global Health: EOT(n= 262, 245) | 51.69 (24.02) | 52.82 (24.48)
  Global Health: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 50.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Global Health: Survival FU 1 (n= 2, 1) | 58.33 (35.36) | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

20. Secondary Outcome: EORTC QLQ-C30 Questionnaire Score: Symptom Subscale
Description: as for outcome 18
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Nausea/Vomiting: Baseline (n= 389, 413) | 8.01 (16.34) | 7.59 (16.35)
  Nausea/Vomiting: C2D1(n= 342, 369) | 11.50 (19.30) | 9.53 (17.25)
  Nausea/Vomiting: C3D1(n= 253, 305) | 7.05 (15.06) | 7.27 (15.32)
  Nausea/Vomiting: C4D1(n= 223, 279) | 7.40 (14.37) | 7.17 (15.50)
  Nausea/Vomiting: C5D1(n= 167, 238) | 6.29 (12.49) | 6.44 (14.54)
  Nausea/Vomiting: C6D1(n= 151, 225) | 6.40 (13.17) | 6.44 (15.16)
  Nausea/Vomiting: C7D1(n= 88, 190) | 6.82 (13.28) | 5.61 (13.74)
  Nausea/Vomiting: C8D1(n= 72, 170) | 6.02 (12.91) | 4.61 (10.57)
  Nausea/Vomiting: C9D1(n= 50, 153) | 3.33 (8.91) | 2.83 (8.06)
  Nausea/Vomiting: C10D1(n= 47, 146) | 2.48 (6.93) | 3.54 (10.02)
  Nausea/Vomiting: C11D1(n= 37, 134) | 3.15 (6.62) | 3.23 (8.54)
  Nausea/Vomiting: C12D1(n= 30, 132) | 3.89 (8.40) | 3.03 (7.66)
  Nausea/Vomiting: C13D1(n= 19, 124) | 4.39 (9.37) | 3.36 (10.19)
  Nausea/Vomiting: C14D1(n= 18, 121) | 4.63 (9.58) | 3.31 (9.03)
  Nausea/Vomiting: C15D1(n= 16, 113) | 1.04 (4.17) | 3.83 (11.14)
  Nausea/Vomiting: C16D1(n= 13, 109) | 5.13 (10.51) | 2.75 (8.64)
  Nausea/Vomiting: C17D1(n= 11, 98) | 9.09 (13.67) | 2.55 (8.06)
  Nausea/Vomiting: C18D1(n= 10, 92) | 6.67 (11.65) | 3.08 (8.88)
  Nausea/Vomiting: C19D1(n= 9, 84) | 3.70 (7.35) | 4.17 (11.53)
  Nausea/Vomiting: C20D1(n= 9, 80) | 5.56 (8.33) | 3.13 (11.28)
  Nausea/Vomiting: C21D1(n= 9, 75) | 1.85 (5.56) | 4.89 (13.08)
  Nausea/Vomiting: C22D1(n= 8, 69) | 6.25 (8.63) | 1.93 (7.31)
  Nausea/Vomiting: C23D1(n= 8, 66) | 6.25 (12.40) | 2.53 (6.69)
  Nausea/Vomiting: C24D1(n= 5, 64) | 0.00 (0.00) | 2.34 (7.19)
  Nausea/Vomiting: C25D1(n= 3, 60) | 0.00 (0.00) | 1.94 (6.21)
  Nausea/Vomiting: C26D1(n= 3, 55) | 0.00 (0.00) | 2.73 (8.34)
  Nausea/Vomiting: C27D1(n= 3, 52) | 0.00 (0.00) | 2.24 (6.62)
  Nausea/Vomiting: C28D1(n= 1, 49) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 1.02 (4.04)
  Nausea/Vomiting: C29D1(n= 2, 40) | 33.33 (47.14) | 1.67 (5.06)
  Nausea/Vomiting: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 1.61 (5.01)
  Nausea/Vomiting: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 2.08 (5.63)
  Nausea/Vomiting: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 1.52 (4.90)
  Nausea/Vomiting: C33D1(n= 0,16) | NA (NA) — Data not reported because no participant was evaluated for this category | 1.04 (4.17)
  Nausea/Vomiting: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 2.38 (8.91)
  Nausea/Vomiting: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 1.39 (4.81)
  Nausea/Vomiting: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.78)
  Nausea/Vomiting: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.67 (9.13)
  Nausea/Vomiting: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Nausea/Vomiting: EOT(n= 266, 245) | 11.65 (20.11) | 10.61 (17.62)
  Nausea/Vomiting: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 16.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Nausea/Vomiting: Survival FU 1 (n= 2, 1) | 50.00 (70.71) | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Pain: Baseline (n= 390, 413) | 29.70 (29.45) | 29.98 (29.72)
  Pain: C2D1(n= 343, 368) | 28.43 (27.24) | 29.30 (29.03)
  Pain: C3D1(n= 256, 305) | 22.59 (24.93) | 24.15 (27.50)
  Pain: C4D1(n= 224, 280) | 21.65 (24.48) | 23.75 (25.84)
  Pain: C5D1(n= 167, 239) | 20.96 (22.55) | 23.22 (25.41)
  Pain: C6D1(n= 151, 225) | 22.41 (21.95) | 21.63 (24.68)
  Pain: C7D1(n= 88, 190) | 21.59 (22.34) | 21.58 (25.30)
  Pain: C8D1(n= 72, 171) | 23.38 (22.49) | 22.03 (24.36)
  Pain: C9D1(n= 50, 153) | 16.33 (20.89) | 19.28 (23.50)
  Pain: C10D1(n= 47, 146) | 14.54 (17.93) | 21.00 (24.61)
  Pain: C11D1(n= 37, 134) | 13.96 (22.05) | 21.27 (26.60)
  Pain: C12D1(n= 30, 132) | 13.33 (21.17) | 18.69 (24.71)
  Pain: C13D1(n= 19, 124) | 16.67 (25.46) | 17.74 (21.23)
  Pain: C14D1(n= 18, 120) | 12.04 (15.97) | 17.64 (22.17)
  Pain: C15D1(n= 16, 113) | 10.42 (17.08) | 17.40 (22.86)
  Pain: C16D1(n= 13, 109) | 21.79 (21.93) | 20.64 (25.25)
  Pain: C17D1(n= 11, 98) | 16.67 (19.72) | 20.41 (25.39)
  Pain: C18D1(n= 10, 92) | 11.67 (22.29) | 20.83 (24.54)
  Pain: C19D1(n= 9, 84) | 14.81 (22.74) | 22.42 (28.16)
  Pain: C20D1(n=9, 80) | 27.78 (31.18) | 20.00 (23.78)
  Pain: C21D1(n= 9, 75) | 14.81 (17.57) | 19.78 (25.95)
  Pain: C22D1(n= 8, 69) | 18.75 (20.77) | 15.22 (19.75)
  Pain: C23D1(n= 8, 66) | 14.58 (27.37) | 16.92 (23.11)
  Pain: C24D1(n=5, 64) | 30.00 (36.13) | 20.05 (25.05)
  Pain: C25D1(n= 3, 60) | 16.67 (28.87) | 18.33 (22.90)
  Pain: C26D1(n= 3, 55) | 22.22 (19.24) | 16.36 (21.87)
  Pain: C27D1(n= 3, 52) | 11.11 (19.24) | 15.06 (20.41)
  Pain: C28D1(n= 1, 49) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 14.29 (18.63)
  Pain: C29D1(n= 2, 40) | 41.67 (58.93) | 13.75 (18.06)
  Pain: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 15.05 (21.24)
  Pain: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 14.58 (21.03)
  Pain: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 16.67 (24.67)
  Pain: C33D1(n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 20.83 (27.55)
  Pain: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 26.19 (27.51)
  Pain: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 22.22 (25.95)
  Pain: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 22.92 (34.43)
  Pain: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 30.00 (34.16)
  Pain: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Pain: EOT (n= 267, 247) | 32.21 (30.36) | 35.43 (31.22)
  Pain: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 16.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Pain: Survival FU-1 (n= 2,1) | 66.67 (47.14) | 83.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Fatigue: Baseline (n= 390, 413) | 37.59 (25.69) | 36.21 (23.92)
  Fatigue: C2D1(n= 343, 369) | 40.52 (25.68) | 39.78 (26.17)
  Fatigue: C3D1(n= 256, 304) | 35.29 (23.97) | 33.90 (23.75)
  Fatigue: C4D1(n= 224, 278) | 35.59 (23.10) | 30.72 (22.57)
  Fatigue: C5D1(n= 167, 238) | 36.03 (22.40) | 30.95 (24.13)
  Fatigue: C6D1(n= 151, 225) | 36.28 (23.40) | 28.89 (22.66)
  Fatigue: C7D1(n= 88, 190) | 34.34 (23.02) | 28.33 (22.15)
  Fatigue: C8D1(n= 72, 170) | 30.86 (24.12) | 27.97 (21.56)
  Fatigue: C9D1(n= 50, 153) | 28.67 (23.45) | 25.78 (21.39)
  Fatigue: C10D1(n= 47, 145) | 29.31 (25.21) | 26.32 (22.27)
  Fatigue: C11D1(n= 37, 134) | 27.63 (25.07) | 25.62 (23.05)
  Fatigue: C12D1(n= 30, 132) | 28.89 (23.99) | 26.60 (23.37)
  Fatigue: C13D1(n= 19, 124) | 22.22 (20.29) | 27.51 (22.73)
  Fatigue: C14D1(n= 18, 121) | 21.60 (16.82) | 26.31 (23.13)
  Fatigue: C15D1(n= 16, 112) | 20.14 (18.24) | 27.73 (22.56)
  Fatigue: C16D1(n= 13, 109) | 21.79 (17.64) | 27.22 (23.35)
  Fatigue: C17D1(n= 11, 98) | 22.22 (12.17) | 27.21 (23.56)
  Fatigue: C18D1(n= 10, 92) | 26.67 (17.53) | 27.29 (24.18)
  Fatigue: C19D1(n= 9, 84) | 22.22 (14.70) | 27.65 (22.85)
  Fatigue: C20D1(n= 9, 80) | 32.10 (30.15) | 25.21 (23.47)
  Fatigue: C21D1(n= 9, 75) | 28.39 (18.52) | 26.44 (23.66)
  Fatigue: C22D1(n= 8, 69) | 33.33 (29.10) | 22.38 (21.77)
  Fatigue: C23D1(n= 8, 66) | 25.00 (24.31) | 24.16 (20.59)
  Fatigue: C24D1(n= 5, 64) | 31.11 (40.37) | 23.78 (18.87)
  Fatigue: C25D1(n= 3, 60) | 11.11 (19.24) | 23.89 (20.94)
  Fatigue: C26D1(n= 3, 55) | 18.52 (16.97) | 28.69 (24.54)
  Fatigue: C27D1(n= 3, 52) | 11.11 (19.24) | 22.65 (19.80)
  Fatigue: C28D1(n= 1, 49) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 22.34 (18.23)
  Fatigue: C29D1(n= 2, 40) | 44.44 (47.14) | 21.11 (18.63)
  Fatigue: C30D1(n= 1, 31) | 22.22 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 23.66 (20.23)
  Fatigue: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 23.15 (20.96)
  Fatigue: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 25.25 (20.63)
  Fatigue: C33D1(n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 29.86 (26.52)
  Fatigue: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 31.75 (24.21)
  Fatigue: C35D1(n= 0, 12) | NA (NA) — Data not reported because no participant was evaluated for this category | 25.00 (21.25)
  Fatigue: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 16.67 (15.71)
  Fatigue: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 24.44 (16.48)
  Fatigue: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 16.67 (7.86)
  Fatigue: EOT(n= 267, 246) | 47.50 (26.72) | 43.07 (28.15)
  Fatigue: Pro Week 6 Pd(n= 0, 1) | NA (NA) — Data not reported because no participant was evaluated for this category | 44.44 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Fatigue: Survival FU-1 (n= 2, 1) | 83.33 (23.57) | 88.89 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

21. Secondary Outcome: EORTC QLQ-LC13 Questionnaire Score: Alopecia
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy experienced during past 1 week. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts. Response range: (1) not at all to (4) very much. Scores for each item were transformed to 0 to 100, where higher symptom score = greater degree of symptoms. Results have been reported for alopecia.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Alopecia: Baseline (n= 384, 405) | 13.89 (27.95) | 14.32 (29.07)
  Alopecia: C2D1(n= 332, 357) | 60.44 (36.66) | 6.63 (16.84)
  Alopecia: C3D1(n= 248, 300) | 56.72 (35.86) | 7.44 (18.89)
  Alopecia: C4D1(n= 219, 270) | 52.36 (35.24) | 7.41 (19.14)
  Alopecia: C5D1(n= 163, 234) | 56.65 (37.25) | 6.41 (16.68)
  Alopecia: C6D1(n= 147, 220) | 54.42 (37.64) | 7.88 (19.34)
  Alopecia: C7D1(n= 87, 186) | 52.11 (39.28) | 5.91 (16.10)
  Alopecia: C8D1(n= 70, 166) | 48.57 (37.94) | 6.63 (17.68)
  Alopecia: C9D1(n= 47, 150) | 48.23 (39.81) | 5.11 (14.83)
  Alopecia: C10D1(n= 45, 142) | 49.63 (39.96) | 3.76 (13.23)
  Alopecia: C11D1(n= 36, 130) | 47.22 (45.34) | 3.08 (11.33)
  Alopecia: C12D1(n= 29, 129) | 36.78 (43.04) | 4.91 (13.88)
  Alopecia: C13D1(n= 19, 121) | 42.11 (41.34) | 6.06 (15.52)
  Alopecia: C14D1(n= 18, 119) | 29.63 (35.95) | 5.60 (14.60)
  Alopecia: C15D1(n= 16, 110) | 33.33 (34.43) | 7.27 (17.12)
  Alopecia: C16D1(n= 12, 105) | 27.78 (31.25) | 7.30 (17.89)
  Alopecia: C17D1(n= 11, 95) | 21.21 (30.81) | 9.47 (19.85)
  Alopecia: C18D1(n= 9, 90) | 22.22 (33.33) | 8.89 (17.16)
  Alopecia: C19D1(n= 8, 81) | 25.00 (34.50) | 10.29 (18.74)
  Alopecia: C20D1(n= 9, 78) | 44.44 (44.10) | 8.55 (15.60)
  Alopecia: C21D1(n= 9, 73) | 22.22 (33.33) | 9.59 (16.18)
  Alopecia: C22D1(n= 7, 67) | 9.52 (16.26) | 9.45 (16.21)
  Alopecia: C23D1(n= 8, 64) | 29.17 (37.53) | 11.46 (18.99)
  Alopecia: C24D1(n= 5, 62) | 13.33 (18.26) | 8.06 (15.61)
  Alopecia: C25D1(n= 2, 58) | 0.00 (0.00) | 9.77 (16.53)
  Alopecia: C26D1(n= 2, 53) | 0.00 (0.00) | 9.43 (16.51)
  Alopecia: C27D1(n= 3, 50) | 33.33 (57.74) | 9.33 (16.55)
  Alopecia: C28D1(n= 2, 46) | 0.00 (0.00) | 6.52 (15.10)
  Alopecia: C29D1(n= 2, 38) | 0.00 (0.00) | 8.77 (20.04)
  Alopecia: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 10.75 (19.98)
  Alopecia: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 9.72 (20.80)
  Alopecia: C32D1(n= 0, 23) | NA (NA) — Data not reported because no participant was evaluated for this category | 7.25 (19.99)
  Alopecia: C33D1(n= 0,16) | NA (NA) — Data not reported because no participant was evaluated for this category | 8.33 (22.77)
  Alopecia: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 9.52 (20.38)
  Alopecia: C35D1(n= 0, 11) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.06 (13.48)
  Alopecia: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.78)
  Alopecia: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.67 (14.91)
  Alopecia: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Alopecia: EOT(n= 261, 243) | 53.51 (38.91) | 6.58 (17.48)
  Alopecia: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 100.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Alopecia: Survival FU 1 (n= 2, 1) | 100.00 (0.00) | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

22. Secondary Outcome: EORTC QLQ-LC13 Questionnaire Score: Coughing
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy experienced during past 1 week. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts. Response range: (1) not at all to (4) very much. Scores for each item were transformed to 0 to 100, where higher symptom score = greater degree of symptoms. Results have been reported for coughing.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Coughing: Baseline (n= 383, 406) | 38.73 (29.64) | 37.27 (27.23)
  Coughing: C2D1(n= 333, 360) | 36.54 (28.04) | 37.50 (28.33)
  Coughing: C3D1(n= 250, 298) | 33.73 (27.46) | 33.89 (24.99)
  Coughing: C4D1(n= 219, 272) | 31.35 (24.13) | 32.48 (25.52)
  Coughing: C5D1(n= 164, 235) | 32.72 (23.49) | 31.35 (25.52)
  Coughing: C6D1(n= 147, 219) | 31.75 (24.78) | 31.05 (24.73)
  Coughing: C7D1(n= 87, 185) | 32.95 (24.64) | 30.99 (25.07)
  Coughing: C8D1(n= 69, 166) | 30.43 (28.43) | 29.12 (25.73)
  Coughing: C9D1(n= 50, 150) | 24.67 (17.57) | 29.11 (24.52)
  Coughing: C10D1(n= 47, 140) | 23.40 (19.55) | 27.86 (22.83)
  Coughing: C11D1(n= 37, 129) | 21.62 (19.59) | 27.39 (23.37)
  Coughing: C12D1(n= 30, 129) | 20.00 (18.77) | 25.06 (23.95)
  Coughing: C13D1(n= 19, 121) | 15.79 (17.10) | 24.79 (23.78)
  Coughing: C14D1(n= 18, 119) | 16.67 (17.15) | 24.37 (22.42)
  Coughing: C15D1(n= 16, 110) | 12.50 (16.67) | 25.76 (23.31)
  Coughing: C16D1(n= 13, 106) | 20.51 (21.68) | 24.53 (22.21)
  Coughing: C17D1(n= 11, 94) | 21.21 (16.82) | 24.82 (23.92)
  Coughing: C18D1(n= 10, 90) | 26.67 (21.08) | 26.30 (24.22)
  Coughing: C19D1(n= 9, 82) | 22.22 (16.67) | 25.61 (26.86)
  Coughing: C20D1(n= 9, 78) | 25.93 (14.70) | 28.21 (26.36)
  Coughing: C21D1(n= 9, 73) | 22.22 (16.67) | 28.77 (27.95)
  Coughing: C22D1(n= 8, 67) | 25.00 (38.83) | 22.89 (23.36)
  Coughing: C23D1(n= 8, 64) | 20.83 (17.25) | 23.44 (26.35)
  Coughing: C24D1(n= 5, 62) | 26.67 (14.91) | 24.73 (23.33)
  Coughing: C25D1(n= 3, 58) | 33.33 (0.00) | 25.86 (23.40)
  Coughing: C26D1(n= 3, 53) | 44.44 (19.25) | 26.41 (24.77)
  Coughing: C27D1(n= 3, 50) | 11.11 (19.24) | 24.67 (22.14)
  Coughing: C28D1(n= 2, 46) | 16.67 (23.57) | 20.29 (20.46)
  Coughing: C29D1(n= 2, 38) | 16.67 (23.57) | 19.30 (22.77)
  Coughing: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 18.28 (20.80)
  Coughing: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 23.61 (25.02)
  Coughing: C32D1(n= 0, 23) | NA (NA) — Data not reported because no participant was evaluated for this category | 26.09 (19.99)
  Coughing: C33D1(n= 0,16) | NA (NA) — Data not reported because no participant was evaluated for this category | 27.08 (32.70)
  Coughing: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 26.19 (29.75)
  Coughing: C35D1(n= 0, 11) | NA (NA) — Data not reported because no participant was evaluated for this category | 21.21 (22.47)
  Coughing: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 25.00 (15.43)
  Coughing: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 26.67 (14.91)
  Coughing: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 33.33 (0.00)
  Coughing: EOT(n= 262, 246) | 35.75 (27.03) | 38.48 (26.95)
  Coughing: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Coughing: Survival FU 1 (n= 2, 1) | 50.00 (23.57) | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

23. Secondary Outcome: EORTC QLQ-LC13 Questionnaire Score: Dysphagia
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy experienced during past 1 week. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts. Response range: (1) not at all to (4) very much. Scores for each item were transformed to 0 to 100, where higher symptom score = greater degree of symptoms. Results have been reported for dysphagia.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Dysphagia: Baseline (n= 387, 406) | 6.20 (17.52) | 5.09 (15.05)
  Dysphagia: C2D1(n= 336, 358) | 10.22 (21.50) | 6.42 (15.75)
  Dysphagia: C3D1(n= 251, 301) | 9.16 (20.87) | 5.43 (14.53)
  Dysphagia: C4D1(n= 217, 272) | 8.60 (19.45) | 5.88 (16.39)
  Dysphagia: C5D1(n= 163, 236) | 6.75 (16.63) | 6.64 (16.79)
  Dysphagia: C6D1(n= 147, 219) | 6.80 (15.58) | 4.72 (13.28)
  Dysphagia: C7D1(n= 87, 187) | 4.21 (11.14) | 5.70 (15.17)
  Dysphagia: C8D1(n=70, 167) | 5.71 (12.65) | 4.79 (12.82)
  Dysphagia: C9D1(n= 50, 151) | 1.33 (6.60) | 4.64 (14.42)
  Dysphagia: C10D1(n= 47, 143) | 1.42 (6.80) | 5.36 (15.14)
  Dysphagia: C11D1(n= 37, 130) | 1.80 (7.64) | 2.82 (11.01)
  Dysphagia: C12D1(n= 29, 129) | 2.30 (8.60) | 3.88 (12.93)
  Dysphagia: C13D1(n= 19, 121) | 0.00 (0.00) | 3.86 (11.54)
  Dysphagia: C14D1(n= 18, 119) | 5.56 (12.78) | 5.04 (13.47)
  Dysphagia: C15D1(n= 16, 110) | 0.00 (0.00) | 3.33 (11.01)
  Dysphagia: C16D1(n= 13, 106) | 0.00 (0.00) | 3.77 (12.45)
  Dysphagia: C17D1(n= 11, 95) | 3.03 (10.05) | 3.86 (13.63)
  Dysphagia: C18D1(n= 10, 90) | 0.00 (0.00) | 4.44 (15.96)
  Dysphagia: C19D1(n= 9, 82) | 3.70 (11.11) | 5.28 (15.24)
  Dysphagia: C20D1(n= 9, 78) | 0.00 (0.00) | 4.70 (12.85)
  Dysphagia: C21D1(n= 9, 73) | 0.00 (0.00) | 5.02 (15.39)
  Dysphagia: C22D1(n= 8, 67) | 0.00 (0.00) | 2.99 (11.21)
  Dysphagia: C23D1(n= 8, 64) | 0.00 (0.00) | 3.65 (12.05)
  Dysphagia: C24D1(n= 5, 62) | 0.00 (0.00) | 4.84 (15.79)
  Dysphagia: C25D1(n= 3, 58) | 0.00 (0.00) | 4.02 (15.39)
  Dysphagia: C26D1(n= 3, 53) | 0.00 (0.00) | 4.40 (13.14)
  Dysphagia: C27D1(n= 3, 50) | 0.00 (0.00) | 2.67 (11.35)
  Dysphagia: C28D1(n= 2, 46) | 0.00 (0.00) | 4.35 (15.09)
  Dysphagia: C29D1(n= 2, 38) | 0.00 (0.00) | 4.39 (13.80)
  Dysphagia: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 5.38 (15.15)
  Dysphagia: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 5.56 (21.23)
  Dysphagia: C32D1(n= 0, 23) | NA (NA) — Data not reported because no participant was evaluated for this category | 7.25 (17.28)
  Dysphagia: C33D1(n= 0,16) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.25 (13.44)
  Dysphagia: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 9.52 (20.38)
  Dysphagia: C35D1(n= 0, 11) | NA (NA) — Data not reported because no participant was evaluated for this category | 3.03 (10.05)
  Dysphagia: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.78)
  Dysphagia: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.67 (14.91)
  Dysphagia: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Dysphagia: EOT(n= 264, 245) | 10.23 (20.77) | 8.98 (18.87)
  Dysphagia: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Dysphagia: Survival FU 1 (n= 2, 1) | 0.00 (0.00) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

24. Secondary Outcome: EORTC QLQ-LC13 Questionnaire Score: Dyspnea
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy experienced during past 1 week. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts. Response range: (1) not at all to (4) very much. Scores for each item were transformed to 0 to 100, where higher symptom score = greater degree of symptoms. Results have been reported for dyspnea.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Dyspnea: Baseline (n= 386, 407) | 28.55 (23.21) | 26.78 (22.43)
  Dyspnea: C2D1(n= 335, 361) | 28.14 (23.48) | 28.79 (23.67)
  Dyspnea: C3D1(n= 252, 301) | 28.13 (22.45) | 25.40 (20.60)
  Dyspnea: C4D1(n= 220, 273) | 27.75 (19.85) | 25.17 (21.14)
  Dyspnea: C5D1(n= 165, 236) | 26.57 (19.61) | 24.72 (19.90)
  Dyspnea: C6D1(n= 148, 221) | 29.69 (21.94) | 24.01 (21.09)
  Dyspnea: C7D1(n= 87, 187) | 25.35 (21.07) | 24.42 (21.23)
  Dyspnea: C8D1(n=70, 167) | 28.02 (24.12) | 24.42 (22.33)
  Dyspnea: C9D1(n= 50, 151) | 26.00 (21.49) | 22.44 (21.87)
  Dyspnea: C10D1(n= 47, 143) | 27.42 (22.56) | 22.18 (21.35)
  Dyspnea: C11D1(n= 37, 130) | 22.67 (19.79) | 20.43 (21.44)
  Dyspnea: C12D1(n= 30, 129) | 22.41 (18.94) | 22.27 (20.47)
  Dyspnea: C13D1(n= 19, 121) | 16.37 (15.87) | 22.22 (21.52)
  Dyspnea: C14D1(n= 18, 119) | 17.90 (12.13) | 22.41 (20.66)
  Dyspnea: C15D1(n= 16, 110) | 15.28 (12.75) | 22.12 (18.71)
  Dyspnea: C16D1(n= 13, 106) | 14.53 (13.13) | 21.91 (20.71)
  Dyspnea: C17D1(n= 10, 95) | 18.89 (14.86) | 23.51 (21.84)
  Dyspnea: C18D1(n= 10, 90) | 20.00 (12.61) | 22.65 (21.97)
  Dyspnea: C19D1(n= 9, 82) | 18.52 (13.61) | 22.09 (20.91)
  Dyspnea: C20D1(n= 9, 78) | 20.37 (15.21) | 22.65 (21.37)
  Dyspnea: C21D1(n= 9, 73) | 19.75 (15.49) | 20.40 (19.69)
  Dyspnea: C22D1(n= 8, 67) | 18.06 (20.52) | 19.90 (17.68)
  Dyspnea: C23D1(n= 8, 64) | 16.67 (13.28) | 21.2 (19.13)
  Dyspnea: C24D1(n= 5, 62) | 20.00 (14.49) | 21.33 (20.94)
  Dyspnea: C25D1(n= 3, 58) | 29.63 (25.66) | 19.73 (18.39)
  Dyspnea: C26D1(n= 3, 53) | 22.22 (11.11) | 21.80 (19.97)
  Dyspnea: C27D1(n= 3, 50) | 18.52 (6.41) | 20.33 (20.87)
  Dyspnea: C28D1(n= 2, 46) | 5.56 (7.86) | 18.36 (17.87)
  Dyspnea: C29D1(n= 2, 38) | 5.56 (7.86) | 19.30 (16.48)
  Dyspnea: C30D1(n= 1, 31) | 11.11 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 17.92 (17.14)
  Dyspnea: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 24.07 (18.73)
  Dyspnea: C32D1(n= 0, 23) | NA (NA) — Data not reported because no participant was evaluated for this category | 24.15 (20.00)
  Dyspnea: C33D1(n= 0,16) | NA (NA) — Data not reported because no participant was evaluated for this category | 25.69 (27.13)
  Dyspnea: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 27.78 (22.96)
  Dyspnea: C35D1(n= 0, 11) | NA (NA) — Data not reported because no participant was evaluated for this category | 26.26 (19.42)
  Dyspnea: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 18.06 (13.20)
  Dyspnea: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 24.44 (4.97)
  Dyspnea: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 16.67 (7.86)
  Dyspnea: EOT(n= 263, 246) | 36.12 (24.82) | 34.51 (26.36)
  Dyspnea: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 22.22 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Dyspnea: Survival FU 1 (n= 2, 1) | 66.67 (15.71) | 44.44 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

25. Secondary Outcome: EORTC QLQ-LC13 Questionnaire Score: Hemoptysis
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy experienced during past 1 week. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts. Response range: (1) not at all to (4) very much. Scores for each item were transformed to 0 to 100, where higher symptom score = greater degree of symptoms. Results have been reported for hemoptysis.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Hemoptysis: Baseline (n= 386, 406) | 4.32 (13.32) | 3.86 (12.12)
  Hemoptysis: C2D1(n= 336, 359) | 4.76 (14.24) | 3.16 (10.97)
  Hemoptysis: C3D1(n= 251, 301) | 4.38 (13.11) | 3.10 (11.12)
  Hemoptysis: C4D1(n= 220, 270) | 2.88 (10.89) | 2.10 (9.94)
  Hemoptysis: C5D1(n= 163, 234) | 1.43 (7.72) | 1.42 (6.76)
  Hemoptysis: C6D1(n= 148, 219) | 1.80 (7.56) | 1.22 (6.27)
  Hemoptysis: C7D1(n= 87, 187) | 1.15 (6.12) | 1.43 (6.76)
  Hemoptysis: C8D1(n=70, 166) | 1.90 (9.64) | 2.41 (10.09)
  Hemoptysis: C9D1(n= 50, 151) | 2.00 (8.00) | 1.77 (7.49)
  Hemoptysis: C10D1(n= 47, 143) | 2.84 (9.40) | 0.70 (4.79)
  Hemoptysis: C11D1(n= 37, 130) | 1.80 (7.64) | 1.03 (5.78)
  Hemoptysis: C12D1(n= 30, 129) | 0.00 (0.00) | 1.03 (5.80)
  Hemoptysis: C13D1(n= 19, 121) | 3.51 (10.51) | 1.10 (5.98)
  Hemoptysis: C14D1(n= 18, 119) | 1.85 (7.86) | 1.68 (7.32)
  Hemoptysis: C15D1(n= 16, 110) | 0.00 (0.00) | 1.82 (10.91)
  Hemoptysis: C16D1(n= 13, 106) | 0.00 (0.00) | 2.83 (10.41)
  Hemoptysis: C17D1(n= 11, 94) | 0.00 (0.00) | 2.84 (12.61)
  Hemoptysis: C18D1(n= 10, 90) | 0.00 (0.00) | 2.96 (12.88)
  Hemoptysis: C19D1(n= 9, 82) | 0.00 (0.00) | 2.03 (12.11)
  Hemoptysis: C20D1(n= 9, 78) | 0.00 (0.00) | 2.56 (12.90)
  Hemoptysis: C21D1(n= 8, 73) | 0.00 (0.00) | 1.83 (7.64)
  Hemoptysis: C22D1(n= 8, 67) | 0.00 (0.00) | 1.99 (9.85)
  Hemoptysis: C23D1(n= 8, 64) | 0.00 (0.00) | 1.04 (5.85)
  Hemoptysis: C24D1(n= 5, 61) | 0.00 (0.00) | 2.73 (11.05)
  Hemoptysis: C25D1(n= 3, 58) | 0.00 (0.00) | 3.45 (13.52)
  Hemoptysis: C26D1(n= 3, 53) | 0.00 (0.00) | 3.77 (14.11)
  Hemoptysis: C27D1(n= 3, 50) | 0.00 (0.00) | 2.00 (8.00)
  Hemoptysis: C28D1(n= 2, 46) | 33.33 (47.14) | 1.45 (6.87)
  Hemoptysis: C29D1(n= 2, 38) | 0.00 (0.00) | 0.88 (5.41)
  Hemoptysis: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 1.08 (5.99)
  Hemoptysis: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 2.78 (9.41)
  Hemoptysis: C32D1(n= 0, 23) | NA (NA) — Data not reported because no participant was evaluated for this category | 2.90 (9.60)
  Hemoptysis: C33D1(n= 0,16) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Hemoptysis: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Hemoptysis: C35D1(n= 0, 11) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Hemoptysis: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.78)
  Hemoptysis: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Hemoptysis: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Hemoptysis: EOT(n= 264, 243) | 5.18 (14.33) | 6.04 (16.60)
  Hemoptysis: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Hemoptysis: Survival FU 1 (n= 2, 1) | 33.33 (47.14) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

26. Secondary Outcome: EORTC QLQ-LC13 Questionnaire Score: Pain in Arm or Shoulder
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy experienced during past 1 week. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts. Response range: (1) not at all to (4) very much. Scores for each item were transformed to 0 to 100, where higher symptom score = greater degree of symptoms. Results have been reported for pain in arm or shoulder.
Time Frame: Day 1 of each treatment Cycle up to EOT (up to approximately 2.25 years); 6 week following PD (up to approximately 2.25 years); survival follow-up-1 (up to approximately 2.25 years) (1 Cycle= 21 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Pain in Arm or Shoulder: Baseline (n= 384, 405) | 20.49 (28.85) | 20.16 (27.09)
  Pain in Arm or Shoulder: C2D1(n= 332, 358) | 19.58 (27.45) | 18.34 (26.56)
  Pain in Arm or Shoulder: C3D1(n= 248, 294) | 17.20 (27.16) | 16.44 (25.50)
  Pain in Arm or Shoulder: C4D1(n= 217, 270) | 14.75 (23.74) | 18.15 (26.57)
  Pain in Arm or Shoulder: C5D1(n= 164, 232) | 16.06 (24.06) | 14.94 (23.76)
  Pain in Arm or Shoulder: C6D1(n= 147, 219) | 15.42 (23.17) | 15.68 (24.37)
  Pain in Arm or Shoulder: C7D1(n= 86, 184) | 14.73 (23.77) | 16.67 (26.31)
  Pain in Arm or Shoulder: C8D1(n=69, 163) | 15.94 (25.95) | 16.77 (25.22)
  Pain in Arm or Shoulder: C9D1(n= 50, 149) | 14.00 (24.36) | 16.78 (25.89)
  Pain in Arm or Shoulder: C10D1(n= 46, 141) | 14.49 (20.67) | 17.73 (27.18)
  Pain in Arm or Shoulder: C11D1(n= 36, 127) | 11.11 (19.52) | 15.49 (26.82)
  Pain in Arm or Shoulder: C12D1(n= 30, 126) | 12.22 (18.54) | 16.93 (26.91)
  Pain in Arm or Shoulder: C13D1(n= 19, 117) | 12.28 (19.91) | 14.81 (22.93)
  Pain in Arm or Shoulder: C14D1(n= 18, 117) | 11.11 (19.80) | 15.67 (22.56)
  Pain in Arm or Shoulder: C15D1(n= 16, 108) | 12.50 (20.64) | 15.74 (24.31)
  Pain in Arm or Shoulder: C16D1(n= 13, 104) | 7.69 (14.62) | 14.10 (23.54)
  Pain in Arm or Shoulder: C17D1(n= 11, 93) | 9.09 (15.57) | 16.49 (25.83)
  Pain in Arm or Shoulder: C18D1(n= 10, 88) | 13.33 (23.31) | 18.18 (25.73)
  Pain in Arm or Shoulder: C19D1(n= 9, 80) | 7.41 (14.70) | 20.83 (29.23)
  Pain in Arm or Shoulder: C20D1(n= 9, 76) | 11.11 (23.57) | 18.42 (25.18)
  Pain in Arm or Shoulder: C21D1(n= 9, 71) | 11.11 (16.67) | 12.68 (19.81)
  Pain in Arm or Shoulder: C22D1(n= 8, 65) | 16.67 (25.20) | 13.33 (21.89)
  Pain in Arm or Shoulder: C23D1(n= 8, 62) | 16.67 (25.20) | 15.05 (22.32)
  Pain in Arm or Shoulder: C24D1(n= 5, 59) | 20.00 (29.81) | 18.08 (24.23)
  Pain in Arm or Shoulder: C25D1(n= 3, 57) | 11.11 (19.24) | 14.62 (21.84)
  Pain in Arm or Shoulder: C26D1(n= 2, 52) | 16.67 (23.57) | 15.38 (22.35)
  Pain in Arm or Shoulder: C27D1(n= 3, 49) | 11.11 (19.24) | 14.97 (23.63)
  Pain in Arm or Shoulder: C28D1(n= 2, 45) | 0.00 (0.00) | 11.85 (19.01)
  Pain in Arm or Shoulder: C29D1(n= 2, 37) | 0.00 (0.00) | 10.81 (22.30)
  Pain in Arm or Shoulder: C30D1(n= 1, 30) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 10.00 (21.71)
  Pain in Arm or Shoulder: C31D1(n= 0, 23) | NA (NA) — Data not reported because no participant was evaluated for this category | 10.14 (21.17)
  Pain in Arm or Shoulder: C32D1(n= 0, 22) | NA (NA) — Data not reported because no participant was evaluated for this category | 13.64 (26.55)
  Pain in Arm or Shoulder: C33D1(n= 0, 15) | NA (NA) — Data not reported because no participant was evaluated for this category | 20.00 (27.60)
  Pain in Arm or Shoulder: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 16.67 (28.49)
  Pain in Arm or Shoulder: C35D1(n= 0, 11) | NA (NA) — Data not reported because no participant was evaluated for this category | 27.27 (32.72)
  Pain in Arm or Shoulder: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 16.67 (35.63)
  Pain in Arm or Shoulder: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 33.33 (47.14)
  Pain in Arm or Shoulder: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Pain in Arm or Shoulder: EOT(n= 264, 242) | 21.72 (30.48) | 23.14 (29.55)
  Pain in Arm or Shoulder: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Pain in Arm or Shoulder: Survival FU 1 (n= 2, 1) | 83.33 (23.57) | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

27. Secondary Outcome: EORTC QLQ-LC13 Questionnaire Score: Pain in Chest
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy experienced during past 1 week. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts. Response range: (1) not at all to (4) very much. Scores for each item were transformed to 0 to 100, where higher symptom score = greater degree of symptoms. Results have been reported for pain in chest.
Time Frame: as for outcome 26
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Pain in Chest: Baseline (n= 385, 403) | 17.92 (25.33) | 19.52 (26.49)
  Pain in Chest: C2D1(n= 332, 356) | 16.67 (24.65) | 15.26 (22.68)
  Pain in Chest: C3D1(n= 249, 296) | 14.59 (21.92) | 15.43 (23.42)
  Pain in Chest: C4D1(n= 217, 268) | 14.44 (22.37) | 14.43 (23.77)
  Pain in Chest: C5D1(n= 164, 233) | 11.99 (18.42) | 12.16 (19.82)
  Pain in Chest: C6D1(n= 145, 217) | 12.18 (19.96) | 12.60 (21.40)
  Pain in Chest: C7D1(n= 86, 184) | 12.40 (19.83) | 11.78 (20.91)
  Pain in Chest: C8D1(n=69, 164) | 10.63 (20.21) | 14.02 (21.52)
  Pain in Chest: C9D1(n= 49, 149) | 7.48 (17.03) | 10.74 (20.96)
  Pain in Chest: C10D1(n= 46, 142) | 5.07 (12.11) | 8.45 (19.62)
  Pain in Chest: C11D1(n= 36, 127) | 3.70 (10.62) | 9.45 (22.18)
  Pain in Chest: C12D1(n= 30, 128) | 3.33 (10.17) | 8.85 (17.49)
  Pain in Chest: C13D1(n= 19, 120) | 3.51 (10.51) | 7.50 (16.99)
  Pain in Chest: C14D1(n= 18, 118) | 5.56 (12.78) | 7.63 (15.96)
  Pain in Chest: C15D1(n= 16, 109) | 6.25 (13.44) | 8.56 (18.37)
  Pain in Chest: C16D1(n= 13, 105) | 5.13 (12.52) | 8.25 (16.53)
  Pain in Chest: C17D1(n= 11, 94) | 0.00 (0.00) | 8.87 (20.84)
  Pain in Chest: C18D1(n= 10, 89) | 6.67 (14.05) | 7.49 (15.69)
  Pain in Chest: C19D1(n= 9, 80) | 7.41 (14.70) | 7.50 (19.10)
  Pain in Chest: C20D1(n= 9, 76) | 3.70 (11.11) | 10.09 (20.38)
  Pain in Chest: C21D1(n= 9, 71) | 0.00 (0.00) | 7.98 (15.39)
  Pain in Chest: C22D1(n= 8, 66) | 4.17 (11.78) | 7.58 (16.33)
  Pain in Chest: C23D1(n= 8, 62) | 4.17 (11.78) | 7.53 (17.51)
  Pain in Chest: C24D1(n= 5, 61) | 0.00 (0.00) | 8.20 (15.70)
  Pain in Chest: C25D1(n= 3, 57) | 0.00 (0.00) | 8.77 (16.09)
  Pain in Chest: C26D1(n= 2, 52) | 0.00 (0.00) | 10.90 (19.49)
  Pain in Chest: C27D1(n= 3, 49) | 11.11 (19.24) | 8.84 (18.97)
  Pain in Chest: C28D1(n= 2, 45) | 0.00 (0.00) | 8.15 (16.14)
  Pain in Chest: C29D1(n= 2, 37) | 0.00 (0.00) | 8.11 (16.49)
  Pain in Chest: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 5.38 (12.46)
  Pain in Chest: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.26)
  Pain in Chest: C32D1(n= 0, 23) | NA (NA) — Data not reported because no participant was evaluated for this category | 13.04 (19.43)
  Pain in Chest: C33D1(n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 14.58 (24.25)
  Pain in Chest: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 14.29 (25.20)
  Pain in Chest: C35D1(n= 0, 11) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.06 (13.48)
  Pain in Chest: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.78)
  Pain in Chest: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.67 (14.91)
  Pain in Chest: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Pain in Chest: EOT(n= 265, 245) | 18.99 (26.35) | 19.46 (26.95)
  Pain in Chest: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Pain in Chest: Survival FU 1 (n= 2, 1) | 50.00 (70.71) | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

28. Secondary Outcome: EORTC QLQ-LC13 Questionnaire Score: Peripheral Neuropathy
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy experienced during past 1 week. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts. Response range: (1) not at all to (4) very much. Scores for each item were transformed to 0 to 100, where higher symptom score = greater degree of symptoms. Results have been reported for peripheral neuropathy.
Time Frame: as for outcome 26
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Peripheral Neuropathy: Baseline (n= 386, 406) | 19.26 (28.94) | 19.21 (27.77)
  Peripheral Neuropathy: C2D1(n= 335, 358) | 25.57 (29.63) | 20.02 (27.21)
  Peripheral Neuropathy: C3D1(n= 250, 300) | 25.60 (29.16) | 17.78 (25.04)
  Peripheral Neuropathy: C4D1(n= 221, 272) | 28.05 (29.94) | 17.77 (25.75)
  Peripheral Neuropathy: C5D1(n= 165, 235) | 29.29 (28.94) | 18.44 (25.97)
  Peripheral Neuropathy: C6D1(n= 147, 221) | 31.97 (30.69) | 17.50 (25.34)
  Peripheral Neuropathy: C7D1(n= 86, 185) | 31.01 (30.59) | 18.02 (25.29)
  Peripheral Neuropathy: C8D1(n=70, 167) | 35.24 (26.55) | 17.56 (25.30)
  Peripheral Neuropathy: C9D1(n= 50, 150) | 36.00 (29.23) | 15.78 (24.02)
  Peripheral Neuropathy: C10D1(n= 47, 143) | 36.17 (30.16) | 18.18 (25.86)
  Peripheral Neuropathy: C11D1(n= 37, 129) | 27.93 (24.23) | 17.05 (24.69)
  Peripheral Neuropathy: C12D1(n= 30, 129) | 30.00 (25.30) | 17.57 (23.96)
  Peripheral Neuropathy: C13D1(n= 19, 121) | 26.32 (21.02) | 17.91 (25.83)
  Peripheral Neuropathy: C14D1(n= 18, 119) | 25.93 (21.56) | 17.09 (23.72)
  Peripheral Neuropathy: C15D1(n= 15, 110) | 24.44 (15.26) | 17.58 (21.99)
  Peripheral Neuropathy: C16D1(n= 13, 105) | 20.51 (16.88) | 17.14 (24.07)
  Peripheral Neuropathy: C17D1(n= 11, 95) | 21.21 (16.82) | 19.30 (26.44)
  Peripheral Neuropathy: C18D1(n= 10, 90) | 23.33 (22.50) | 18.15 (26.52)
  Peripheral Neuropathy: C19D1(n= 9, 82) | 14.81 (17.57) | 20.33 (26.06)
  Peripheral Neuropathy: C20D1(n= 9, 78) | 22.22 (23.57) | 17.52 (26.17)
  Peripheral Neuropathy: C21D1(n= 9, 73) | 29.63 (20.03) | 18.72 (25.45)
  Peripheral Neuropathy: C22D1(n= 7, 66) | 23.81 (16.26) | 15.66 (23.55)
  Peripheral Neuropathy: C23D1(n= 8, 64) | 16.67 (17.82) | 20.31 (22.71)
  Peripheral Neuropathy: C24D1(n= 5, 62) | 13.33 (18.26) | 20.43 (22.87)
  Peripheral Neuropathy: C25D1(n= 3, 58) | 11.11 (19.24) | 18.39 (20.87)
  Peripheral Neuropathy: C26D1(n= 2, 53) | 16.67 (23.57) | 20.13 (25.60)
  Peripheral Neuropathy: C27D1(n= 3, 50) | 11.11 (19.24) | 19.33 (24.36)
  Peripheral Neuropathy: C28D1(n= 2, 46) | 0.00 (0.00) | 19.57 (22.85)
  Peripheral Neuropathy: C29D1(n= 2, 38) | 0.00 (0.00) | 19.30 (22.77)
  Peripheral Neuropathy: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 20.43 (28.12)
  Peripheral Neuropathy: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 23.61 (26.88)
  Peripheral Neuropathy: C32D1(n= 0, 23) | NA (NA) — Data not reported because no participant was evaluated for this category | 18.84 (22.08)
  Peripheral Neuropathy: C33D1(n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 22.92 (20.07)
  Peripheral Neuropathy: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 19.05 (21.54)
  Peripheral Neuropathy: C35D1(n= 0, 11) | NA (NA) — Data not reported because no participant was evaluated for this category | 15.15 (17.41)
  Peripheral Neuropathy: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 8.33 (15.43)
  Peripheral Neuropathy: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 26.67 (27.89)
  Peripheral Neuropathy: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 16.67 (23.57)
  Peripheral Neuropathy: EOT(n= 262, 244) | 31.81 (31.53) | 19.54 (27.32)
  Peripheral Neuropathy: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Peripheral Neuropathy: Survival FU 1 (n= 2, 1) | 50.00 (23.57) | 33.33 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

29. Secondary Outcome: EORTC QLQ-LC13 Questionnaire Score: Pain in Other Parts
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy experienced during past 1 week. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts. Response range: (1) not at all to (4) very much. Scores for each item were transformed to 0 to 100, where higher symptom score = greater degree of symptoms. Results have been reported for pain in other parts.
Time Frame: as for outcome 26
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Pain in Other Parts: Baseline (n= 373, 402) | 27.52 (30.41) | 27.94 (31.52)
  Pain in Other Parts: C2D1(n= 320, 347) | 29.58 (30.44) | 27.76 (30.53)
  Pain in Other Parts: C3D1(n= 239, 286) | 22.87 (27.79) | 25.87 (29.79)
  Pain in Other Parts: C4D1(n= 211, 263) | 21.48 (26.86) | 23.45 (26.92)
  Pain in Other Parts: C5D1(n= 154, 230) | 21.21 (26.63) | 22.32 (27.24)
  Pain in Other Parts: C6D1(n= 139, 214) | 22.78 (25.39) | 21.50 (27.88)
  Pain in Other Parts: C7D1(n= 81, 180) | 23.05 (28.21) | 24.63 (29.56)
  Pain in Other Parts: C8D1(n=65, 158) | 24.10 (28.57) | 18.35 (24.54)
  Pain in Other Parts: C9D1(n= 44, 135) | 18.18 (28.26) | 21.48 (28.35)
  Pain in Other Parts: C10D1(n= 44, 136) | 15.15 (23.24) | 21.57 (28.84)
  Pain in Other Parts: C11D1(n= 34, 123) | 14.71 (23.49) | 20.05 (27.90)
  Pain in Other Parts: C12D1(n= 26, 122) | 8.97 (17.78) | 16.67 (25.80)
  Pain in Other Parts: C13D1(n= 17, 113) | 17.65 (23.91) | 19.76 (25.05)
  Pain in Other Parts: C14D1(n= 18, 115) | 18.52 (23.49) | 22.03 (29.58)
  Pain in Other Parts: C15D1(n= 15, 106) | 6.67 (13.80) | 19.18 (25.18)
  Pain in Other Parts: C16D1(n= 13, 105) | 20.51 (21.68) | 21.90 (26.89)
  Pain in Other Parts: C17D1(n= 11, 93) | 15.15 (22.92) | 22.22 (27.51)
  Pain in Other Parts: C18D1(n= 10, 89) | 13.33 (23.31) | 22.10 (27.50)
  Pain in Other Parts: C19D1(n= 9, 80) | 18.52 (24.22) | 24.58 (29.88)
  Pain in Other Parts: C20D1(n= 9, 74) | 25.93 (36.43) | 21.17 (27.90)
  Pain in Other Parts: C21D1(n= 8, 69) | 12.50 (17.25) | 21.26 (31.30)
  Pain in Other Parts: C22D1(n= 8, 62) | 20.83 (24.80) | 18.82 (25.34)
  Pain in Other Parts: C23D1(n= 8, 62) | 20.83 (30.54) | 18.82 (23.86)
  Pain in Other Parts: C24D1(n= 5, 61) | 26.67 (43.46) | 19.67 (28.14)
  Pain in Other Parts: C25D1(n= 3, 55) | 11.11 (19.24) | 16.97 (26.35)
  Pain in Other Parts: C26D1(n= 2, 50) | 16.67 (23.57) | 18.67 (26.22)
  Pain in Other Parts: C27D1(n= 3, 49) | 11.11 (19.24) | 14.29 (21.52)
  Pain in Other Parts: C28D1(n= 2, 44) | 0.00 (0.00) | 15.15 (25.37)
  Pain in Other Parts: C29D1(n= 2, 36) | 0.00 (0.00) | 21.30 (26.61)
  Pain in Other Parts: C30D1(n= 1, 30) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 16.67 (30.01)
  Pain in Other Parts: C31D1(n= 0, 23) | NA (NA) — Data not reported because no participant was evaluated for this category | 11.59 (21.58)
  Pain in Other Parts: C32D1(n= 0, 23) | NA (NA) — Data not reported because no participant was evaluated for this category | 20.29 (27.96)
  Pain in Other Parts: C33D1(n= 0, 15) | NA (NA) — Data not reported because no participant was evaluated for this category | 11.11 (27.22)
  Pain in Other Parts: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 30.95 (33.24)
  Pain in Other Parts: C35D1(n= 0, 10) | NA (NA) — Data not reported because no participant was evaluated for this category | 26.67 (34.43)
  Pain in Other Parts: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 20.83 (35.36)
  Pain in Other Parts: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 33.33 (40.82)
  Pain in Other Parts: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Pain in Other Parts: EOT(n= 250, 226) | 30.80 (32.97) | 32.01 (33.89)
  Pain in Other Parts: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Pain in Other Parts: Survival FU 1 (n= 2, 1) | 83.33 (23.57) | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

30. Secondary Outcome: EORTC QLQ-LC13 Questionnaire Score: Sore Mouth
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy experienced during past 1 week. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts. Response range: (1) not at all to (4) very much. Scores for each item were transformed to 0 to 100, where higher symptom score = greater degree of symptoms. Results have been reported for sore mouth.
Time Frame: as for outcome 26
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 425 | 425
Units on a scale
  Sore Mouth: Baseline (n= 387, 404) | 5.68 (16.34) | 4.95 (15.32)
  Sore Mouth: C2D1(n= 335, 357) | 15.52 (25.75) | 7.10 (18.17)
  Sore Mouth: C3D1(n= 252, 297) | 14.29 (23.59) | 5.61 (14.18)
  Sore Mouth: C4D1(n= 219, 270) | 14.00 (22.95) | 4.81 (13.99)
  Sore Mouth: C5D1(n= 165, 234) | 11.31 (19.65) | 4.27 (13.49)
  Sore Mouth: C6D1(n= 148, 218) | 13.29 (23.24) | 4.13 (13.89)
  Sore Mouth: C7D1(n= 87, 185) | 9.20 (20.77) | 5.59 (15.50)
  Sore Mouth: C8D1(n=70, 166) | 8.57 (16.73) | 5.02 (14.96)
  Sore Mouth: C9D1(n= 50, 151) | 6.00 (17.42) | 3.09 (14.06)
  Sore Mouth: C10D1(n= 47, 143) | 7.09 (15.44) | 3.96 (14.53)
  Sore Mouth: C11D1(n= 37, 130) | 4.50 (13.97) | 3.33 (12.35)
  Sore Mouth: C12D1(n= 30, 129) | 2.22 (8.46) | 4.65 (14.87)
  Sore Mouth: C13D1(n= 19, 121) | 1.75 (7.65) | 5.23 (15.52)
  Sore Mouth: C14D1(n= 18, 119) | 3.70 (10.78) | 5.32 (15.64)
  Sore Mouth: C15D1(n= 15, 110) | 0.00 (0.00) | 4.24 (13.63)
  Sore Mouth: C16D1(n= 13, 106) | 0.00 (0.00) | 3.77 (16.15)
  Sore Mouth: C17D1(n= 11, 95) | 3.03 (10.05) | 6.32 (17.73)
  Sore Mouth: C18D1(n= 10, 90) | 3.33 (10.54) | 3.70 (11.66)
  Sore Mouth: C19D1(n= 9, 82) | 0.00 (0.00) | 4.47 (12.57)
  Sore Mouth: C20D1(n= 9, 78) | 0.00 (0.00) | 5.56 (15.59)
  Sore Mouth: C21D1(n= 9, 73) | 0.00 (0.00) | 7.76 (17.14)
  Sore Mouth: C22D1(n= 8, 67) | 4.17 (11.78) | 6.47 (17.64)
  Sore Mouth: C23D1(n= 8, 64) | 4.17 (11.78) | 6.25 (16.67)
  Sore Mouth: C24D1(n= 5, 62) | 0.00 (0.00) | 5.38 (13.75)
  Sore Mouth: C25D1(n= 3, 57) | 0.00 (0.00) | 3.51 (10.32)
  Sore Mouth: C26D1(n= 3, 53) | 0.00 (0.00) | 6.92 (13.65)
  Sore Mouth: C27D1(n= 3, 50) | 0.00 (0.00) | 4.00 (10.94)
  Sore Mouth: C28D1(n= 2, 46) | 0.00 (0.00) | 4.35 (11.35)
  Sore Mouth: C29D1(n= 2, 38) | 0.00 (0.00) | 3.51 (10.37)
  Sore Mouth: C30D1(n= 1, 31) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. | 4.30 (11.36)
  Sore Mouth: C31D1(n= 0, 24) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.26)
  Sore Mouth: C32D1(n= 0, 23) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.35 (11.48)
  Sore Mouth: C33D1(n= 0, 16) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.39)
  Sore Mouth: C34D1(n= 0, 14) | NA (NA) — Data not reported because no participant was evaluated for this category | 9.52 (15.63)
  Sore Mouth: C35D1(n= 0, 11) | NA (NA) — Data not reported because no participant was evaluated for this category | 6.06 (13.48)
  Sore Mouth: C36D1(n= 0, 8) | NA (NA) — Data not reported because no participant was evaluated for this category | 4.17 (11.78)
  Sore Mouth: C37D1(n= 0, 5) | NA (NA) — Data not reported because no participant was evaluated for this category | 13.33 (29.81)
  Sore Mouth: C38D1(n= 0, 2) | NA (NA) — Data not reported because no participant was evaluated for this category | 0.00 (0.00)
  Sore Mouth: EOT(n= 265, 243) | 11.57 (22.85) | 7.00 (17.18)
  Sore Mouth: Pro Week 6 Pd(n= 0,1) | NA (NA) — Data not reported because no participant was evaluated for this category | 66.67 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Sore Mouth: Survival FU 1 (n= 2, 1) | 16.67 (23.57) | 0.00 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.

31. Primary Outcome: OS: SP-ITT
Description: as for outcome 3
Time Frame: Baseline until death due to any cause (up to approximately 2.87 years)
Population: Secondary population (SP) ITT analysis set included all 1225 randomized participants regardless of whether they received any study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 612 | 613
Months | 9.8 [8.8 to 11.3] | 13.3 [11.3 to 14.9]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0012, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.70 to 0.92]

32. Primary Outcome: OS: TC1/2/3 Or IC1/2/3 Subgroup of SP
Description: as for outcome 3
Time Frame: Baseline until death from any cause (approximately 2.87 years)
Population: TC1/2/3 Or IC1/2/3 Subgroup of SP.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 337 | 347
Months | 10.8 [9.3 to 12.0] | 14.3 [12.4 to 16.7]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0045, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.64 to 0.92]

33. Primary Outcome: OS: TC2/3 or IC2/3 Subgroup of SP
Description: as for outcome 3
Time Frame: Baseline until death due to any cause (up to approximately 2.87 years)
Population: TC2/3 or IC2/3 Subgroup of SP.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 182 | 168
Months | 11.4 [9.3 to 12.9] | 16.6 [13.6 to 20.1]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0012, Log Rank; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.49 to 0.84]

34. Primary Outcome: OS: TC3 or IC3 Subgroup of SP
Description: as for outcome 3
Time Frame: Baseline until death due to any cause (up to approximately 2.87 years)
Population: TC3 or IC3 Subgroup of SP.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 85 | 89
Months | 9.7 [7.9 to 11.6] | 20.5 [16.8 to 30.2]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.30 to 0.68]

35. Secondary Outcome: PFS as Determined by Investigator Using RECIST v1.1: SP-ITT
Description: as for outcome 7
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 2.87 years)
Population: SP-ITT analysis set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 612 | 613
Months | 3.8 [3.3 to 4.1] | 2.7 [2.4 to 2.9]
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; Test type: Superiority or Other; p = 0.4981, Log Rank; Stratified Hazard Ratio = 0.96, 95% CI 2-sided [0.85 to 1.08]

36. Secondary Outcome: Percentage of Participants With Objective Response as Determined Using RECIST v1.1: SP-ITT
Description: as for outcome 9
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 2.87 years)
Population: SP-ITT analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 612 | 613
Percentage of Participants | 11.8 [9.32 to 14.59] | 13.7 [11.08 to 16.68]

37. Secondary Outcome: DOR as Determined by Investigator Using RECIST v1.1: SP ITT
Description: as for outcome 11
Time Frame: From first objective response of CR or PR to PD or death due to any cause, whichever occurred first (up to approximately 2.87 years)
Population: The SP-ITT analysis set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Atezolizumab
Number analyzed (Participants) | 72 | 84
Months | 6.3 [5.5 to 7.6] | 23.9 [12.8 to NA] — Data not reported because the upper limit of confidence interval (CI) was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Docetaxel vs Atezolizumab; Test type: Superiority or Other; Unstratified Hazard Ratio = 0.32, 95% CI 2-sided [0.21 to 0.48]

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 5.28 years.
Description: Safety evaluable population included all randomized participants who received any dose of study drug. Analysis was performed according to actual treatment received. One participant randomized to docetaxel received atezolizumab and hence included in atezolizumab arm.
Arm/Group | Docetaxel | Atezolizumab
Serious Adverse Events (participants affected / at risk) | 180/578 | 200/609
Other Adverse Events (participants affected / at risk) | 535/578 | 541/609
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=578) | Atezolizumab (N=609)
Anaemia (Blood and lymphatic system disorders) | 7 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 37 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 2
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 3
Pericarditis (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Oesophageal fistula (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1
Asthenia (General disorders) | 3 | 3
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 2
General physical health deterioration (General disorders) | 0 | 2
Generalised oedema (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 8 | 9
Sudden death (General disorders) | 2 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 2
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 3
Abdominal sepsis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 2 | 0
Encephalitis (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gastrointestinal fungal infection (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 3 | 3
Lung infection (Infections and infestations) | 3 | 3
Meningitis (Infections and infestations) | 0 | 3
Neutropenic sepsis (Infections and infestations) | 2 | 0
Paronychia (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 2
Pleural infection (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 34 | 20
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 4 | 8
Sepsis (Infections and infestations) | 2 | 5
Septic shock (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 5 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 3
Syncope (Nervous system disorders) | 3 | 1
Confusional state (Psychiatric disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Henoch-Schonlein purpura nephritis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Pleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 3
Superior vena cava syndrome (Vascular disorders) | 1 | 3
Thrombosis (Vascular disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Mental status change (Psychiatric disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=578) | Atezolizumab (N=609)
Anaemia (Blood and lymphatic system disorders) | 130 | 71
Neutropenia (Blood and lymphatic system disorders) | 88 | 12
Lacrimation increased (Eye disorders) | 33 | 6
Abdominal pain (Gastrointestinal disorders) | 33 | 23
Constipation (Gastrointestinal disorders) | 82 | 111
Diarrhoea (Gastrointestinal disorders) | 138 | 100
Nausea (Gastrointestinal disorders) | 131 | 110
Stomatitis (Gastrointestinal disorders) | 62 | 21
Vomiting (Gastrointestinal disorders) | 61 | 75
Asthenia (General disorders) | 113 | 117
Chest pain (General disorders) | 25 | 55
Fatigue (General disorders) | 206 | 165
Influenza like illness (General disorders) | 14 | 35
Malaise (General disorders) | 29 | 15
Mucosal inflammation (General disorders) | 41 | 9
Oedema peripheral (General disorders) | 82 | 55
Pyrexia (General disorders) | 70 | 108
Nasopharyngitis (Infections and infestations) | 21 | 39
Upper respiratory tract infection (Infections and infestations) | 15 | 41
Urinary tract infection (Infections and infestations) | 30 | 22
Alanine aminotransferase increased (Investigations) | 14 | 36
Aspartate aminotransferase increased (Investigations) | 12 | 42
Neutrophil count decreased (Investigations) | 50 | 3
Weight decreased (Investigations) | 30 | 56
Decreased appetite (Metabolism and nutrition disorders) | 135 | 150
Arthralgia (Musculoskeletal and connective tissue disorders) | 59 | 80
Back pain (Musculoskeletal and connective tissue disorders) | 41 | 70
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 24 | 69
Myalgia (Musculoskeletal and connective tissue disorders) | 90 | 44
Pain in extremity (Musculoskeletal and connective tissue disorders) | 38 | 56
Dizziness (Nervous system disorders) | 32 | 48
Dysgeusia (Nervous system disorders) | 48 | 18
Headache (Nervous system disorders) | 46 | 62
Neuropathy peripheral (Nervous system disorders) | 65 | 27
Paraesthesia (Nervous system disorders) | 45 | 23
Peripheral sensory neuropathy (Nervous system disorders) | 43 | 5
Depression (Psychiatric disorders) | 6 | 31
Insomnia (Psychiatric disorders) | 43 | 56
Cough (Respiratory, thoracic and mediastinal disorders) | 107 | 146
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 108 | 117
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 28 | 40
Alopecia (Skin and subcutaneous tissue disorders) | 205 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 34 | 30
Nail disorder (Skin and subcutaneous tissue disorders) | 30 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 57
Rash (Skin and subcutaneous tissue disorders) | 51 | 65
Bronchitis (Infections and infestations) | 24 | 34
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 33
Productive cough (Respiratory, thoracic and mediastinal disorders) | 21 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.